CLINICAL TRIAL: NCT02960438
Title: A Dose Response Study of E6011 in Subjects With Rheumatoid Arthritis Inadequately Responding to Methotrexate
Brief Title: A Dose Response Study of E6011 in Participants With Rheumatoid Arthritis Inadequately Responding to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E6011-J081-201
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Rheumatoid Arthritis
Keywords: E6011; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- E6011 100 milligrams (mg) (Experimental): In the Treatment Phase, E6011 100 mg will be subcutaneously administered at Weeks 0, 1, and 2, and then every 2 weeks up to Week 22. In the Extension Phase, E6011 200 mg will be subcutaneously administered every 2 weeks until Week 102.
  Interventions: Drug: E6011
- E6011 200 mg (Experimental): In the Treatment Phase, E6011 200 mg will be subcutaneously administered at Weeks 0, 1, and 2, and then every 2 weeks up to Week 22. In the Extension Phase, E6011 200 mg will be subcutaneously administered every 2 weeks until Week 102.
  Interventions: Drug: E6011
- E6011 400 mg (Experimental): In the Treatment Phase, E6011 400 mg will be subcutaneously administered at Weeks 0, 1, 2, 4, 6, 8, and 10, and then E6011 200 mg will be subcutaneously administered every 2 weeks up to Week 22. In the Extension Phase, E6011 200 mg will be subcutaneously administered every 2 weeks until Week 102.
  Interventions: Drug: E6011
- Placebo (Placebo Comparator): In the Treatment Phase, placebo will be subcutaneously administered at Weeks 0, 1, and 2, and then every 2 weeks up to Week 22. In the Extension Phase, E6011 200 mg will be subcutaneously administered every 2 weeks until Week 102.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6011 — subcutaneous administration
  Arms: E6011 100 milligrams (mg); E6011 200 mg; E6011 400 mg
Drug: Placebo — subcutaneous administration
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel-group comparison study in rheumatoid arthritis participants inadequately responding to methotrexate.

ELIGIBILITY:
Inclusion Criteria

* Aged greater than or equal to (>=) 18 and less than (<)75 years old at the time of informed consent
* Diagnosed with rheumatoid arthritis (RA) under the 1987 American College of Rheumatology (ACR) or 2010 ACR/European League Against Rheumatism (EULAR) criteria >=12 weeks before informed consent
* Received methotrexate (MTX) treatment at 6 to 16 milligram (mg)/week for >=12 weeks before screening and presented ≥6 tender joints (out of 68 joints) and >=6 swollen joints (out of 66 joints) in the Screening and Observation Phases
* Can continue stable dose regimen of MTX at 6 to 16 mg/week from 4 weeks before starting the study treatment until completion of the Extension Phase (or until study discontinuation)
* C-reactive protein (CRP) level >=0.6 mg/deciliter (dL) or erythrocyte sedimentation rate (ESR) >=28 millimeters per hour (mm/hr) in the Screening Phase
* Erosions at >=3 sites in radiographic image in the Screening Phase, or those with erosions at >=1 site and either positive for rheumatoid factor (RF) or anti-cyclic citrullinated peptide (CCP) antibody in the Screening Phase
* Weighs >=30 kilograms (kg) and ≤100 kg in the Screening Phase
* Has voluntarily consented, in writing, to participate in this study. If a participant is below the age of 20, also consented, in writing, by a legally acceptable representative.
* Has been thoroughly briefed on the conditions for participation in the study, is able to understand, and is willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Any history or complication of inflammatory arthritic disorder other than RA or Sjogren's syndrome
* Meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class IV in the Screening Phase
* Received immunoglobulin preparations or blood products within 24 weeks before starting the study treatment
* Received a live vaccine within 12 weeks before starting the study treatment, or is planning to receive
* Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, or renal disease) that could affect the participant's safety or interfere with the study assessments in the opinion of the investigator or subinvestigator
* Complication of uncontrolled disorders such as acute cardiac infarction, unstable angina, brain infarct, or symptomatic intracerebral hemorrhage
* History of severe allergy (shock or anaphylactoid symptoms)
* History or current clinical condition of malignant tumor, lymphoma, leukemia, or lymphoproliferative disease, except for skin carcinoma (epithelial carcinoma or basal cell carcinoma) and cervix carcinoma which has completely excised and without metastasis or recurrence for more than 5 years before informed consent
* Immunodeficiency or history of human immunodeficiency virus (HIV) infection
* Infection requiring hospitalization or intravenous administration of antibiotics or disease requiring administration of antivirus drugs (example, herpes zoster) within 4 weeks before starting the study treatment
* History of tuberculosis or current complication of active tuberculosis
* History of clinically important vasculitis
* Tested positive for any of the following in the Screening Phase: HIV, hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B virus core antibody (HBc antibody), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C virus antibody (HCV antibody), human T-lymphotrophic virus Type I antibody (HTLV-1 antibody), or syphilis
* Positive in tuberculosis test (QuantiFERON®TB Gold Test or T-SPOT®.TB Test) in the Screening Phase
* Findings indicating a history of tuberculosis on chest x-ray in the Screening Phase
* Neurological findings such as paralysis, visual impairment, or language disorder in the Screening Phase
* Demonstrated prolonged QTcF interval (>450 milliseconds [ms]) in repeated electrocardiogram examinations
* Females of childbearing potential who have a positive pregnancy test in the Screening or Observation Phase or are breastfeeding
* Females of childbearing potential who:

  * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation
  * Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from being sexually active during the study period or for 28 days after study drug discontinuation
  * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]).
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 28 days after study drug discontinuation.
* Scheduled for surgery during the study
* Currently enrolled in another clinical study or used any investigational drug or device within 28 days (or 5* the half-life, whichever is longer) before informed consent
* Has been treated with E6011 or any biologics for use in RA that has not been approved
* Use of a psychotropic agent as recreational purpose other than therapeutic purpose
* Any history of a medical condition or a concomitant medical condition that in the opinion of the investigator or subinvestigator would compromise the participant's ability to safely complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- Japan (90):
  - Eisai Trial Site #1, Nagoya, Aichi-ken
  - Eisai Trial Site #2, Nagoya, Aichi-ken
  - Eisai Trial Site #3, Nagoya, Aichi-ken
  - Eisai Trial Site #4, Nagoya, Aichi-ken
  - Eisai Trial Site #1, Toyohashi, Aichi-ken
  - Eisai Trial Site #1, Toyota, Aichi-ken
  - Eisai Trial Site #1, Funabashi, Chiba
  - Eisai Trial Site #1, Matsuyama, Ehime
  - Eisai Trial Site #1, Iizuka, Fukuoka
  - Eisai Trial Site #1, Kitakyushu, Fukuoka
  - Eisai Trial Site #1, Kurume, Fukuoka
  - Eisai Trial Site #2, Kurume, Fukuoka
  - Eisai Trial Site #1, Takasaki, Gunma
  - Eisai Trial Site #2, Takasaki, Gunma
  - Eisai Trial Site #1, Asahikawa, Hokkaido
  - Eisai Trial Site #1, Hakodate, Hokkaido
  - Eisai Trial Site #1, Kushiro, Hokkaido
  - Eisai Trial Site #1, Sapporo, Hokkaido
  - Eisai Trial Site #2, Sapporo, Hokkaido
  - Eisai Trial Site #3, Sapporo, Hokkaido
  - Eisai Trial Site #1, Tomakomai, Hokkaido
  - Eisai Trial Site #1, Kobe, Hyōgo
  - Eisai Trial Site #1, Takarazuka, Hyōgo
  - Eisai Trial Site #1, Hitachi, Ibaraki
  - Eisai Trial Site #1, Hitachi-Naka, Ibaraki
  - Eisai Trial Site #1, Kasama, Ibaraki
  - Eisai Trial Site #1, Komatsu, Ishikawa-ken
  - Eisai Trial Site #1, Morioka, Iwate
  - Eisai Trial Site #1, Kirishima, Kagoshima-ken
  - Eisai Trial Site #1, Yokohama, Kanagawa
  - Eisai Trial Site #2, Yokohama, Kanagawa
  - Eisai Trial Site #1, Yamaga, Kumamoto
  - Eisai Trial Site #1, Yokkaichi, Mie-ken
  - Eisai Trial Site #1, Ōsaki, Miyagi
  - Eisai Trial Site #1, Sendai, Miyagi
  - Eisai Trial Site #2, Sendai, Miyagi
  - Eisai Trial Site #1, Hyūga, Miyazaki
  - Eisai Trial site #2, Hyūga, Miyazaki
  - Eisai Trial Site #1, Matsumoto, Nagano
  - Eisai Trial Site #1, Isahaya, Nagasaki
  - Eisai Trial Site #1, Ōmura, Nagasaki
  - Eisai Trial Site #1, Sasebo, Nagasaki
  - Eisai Trial Site #1, Nagaoka, Niigata
  - Eisai Trial Site #1, Shibata, Niigata
  - Eisai Trial Site #1, Beppu, Oita Prefecture
  - Eisai Trial Site #1, Tomigusuku, Okinawa
  - Eisai Trial Site #1, Kawachi-Nagano, Osaka
  - Eisai Trial Site #1, Ureshino, Saga-ken
  - Eisai Trial Site #1, Hiki, Saitama
  - Eisai Trial Site #1, Kawagoe, Saitama
  - Eisai Trial Site #1, Kawaguchi, Saitama
  - Eisai Trial Site #1, Tokorozawa, Saitama
  - Eisai Trial Site #1, Hamamatsu, Shizuoka
  - Eisai Trial Site #1, Shimotsuke, Tochigi
  - Eisai Trial Site #1, Bunkyo, Tokyo
  - Eisai Trial Site #1, Chūō, Tokyo
  - Eisai Trial Site #1, Fuchū, Tokyo
  - Eisai Trial Site #1, Meguro City, Tokyo
  - Eisai Trial Site #1, Musashino, Tokyo
  - Eisai Trial Site #1, Nakano City, Tokyo
  - Eisai Trial Site #1, Ōme, Tokyo
  - Eisai Trial Site #1, Ōta-ku, Tokyo
  - Eisai Trial Site #1, Setagaya City, Tokyo
  - Eisai Trial Site #1, Shinjuku, Tokyo
  - Eisai Trial Site #2, Shinjuku, Tokyo
  - Eisai Trial Site #1, tabashi City, Tokyo
  - Eisai Trial Site #1, Takaoka, Toyama
  - Eisai Trial Site #1, Nishimuro, Wakayama
  - Eisai Trial Site #1, Shimonoseki, Yamaguchi
  - Eisai Trial Site #2, Shimonoseki, Yamaguchi
  - Eisai Trial Site #1, Fukui
  - Eisai Trial Site #2, Fukuoka
  - Eisai Trial Site #1, Gifu
  - Eisai Trial Site #1, Hiroshima
  - Eisai Trial Site #2, Hiroshima
  - Eisai Trial Site #3, Hiroshima
  - Eisai Trial Site #1, Kagoshima
  - Eisai Trial Site #2, Kagoshima
  - Eisai Trial Site #3, Kagoshima
  - Eisai Trial Site #1, Kochi
  - Eisai Trial Site #2, Kumamoto
  - Eisai Trial Site #1, Miyagi
  - Eisai Trial Site #1, Miyazaki
  - Eisai Trial Site #1, Nagano
  - Eisai Trial Site #1, Nagasaki
  - Eisai Trial Site #2, Nagasaki
  - Eisai Trial Site #3, Nagasaki
  - Eisai Trial Site #1, Ōita
  - Eisai Trial Site #1, Saitama
  - Eisai Trial Site #1, Shizuoka

REFERENCES:
- [Derived] Tanaka Y, Takeuchi T, Yamanaka H, Nanki T, Umehara H, Yasuda N, Tago F, Kitahara Y, Kawakubo M, Torii K, Hojo S, Kawano T, Imai T. Efficacy and Safety of E6011, an Anti-Fractalkine Monoclonal Antibody, in Patients With Active Rheumatoid Arthritis With Inadequate Response to Methotrexate: Results of a Randomized, Double-Blind, Placebo-Controlled Phase II Study. Arthritis Rheumatol. 2021 Apr;73(4):587-595. doi: 10.1002/art.41555. Epub 2021 Feb 18. PMID 33038062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 91 investigative sites in Japan from 20 October 2016 to 17 September 2019.
Pre-assignment Details: A total of 273 participants were screened and enrolled (signed informed consent form), of which 79 were screen failures, and 194 were randomized out which 190 received study treatment.
Groups:
- Placebo: During Treatment Phase, participants received E6011-matched placebo, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase and received E6011 200 milligram (mg), infusion, subcutaneously, every 2 weeks until Week 102.
- E6011 100 mg: During Treatment Phase, participants received E6011 100 mg, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
- E6011 200 mg: During Treatment Phase, participants received E6011 200 mg, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
- E6011 400/200 mg: During Treatment Phase, participants received E6011 400 mg, infusion, subcutaneously, at Weeks 0, 1, 4, 6, 8, 10 and then E6011 200 mg, infusion, subcutaneously, every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
Period: Treatment Phase (Double-blind): 24 Weeks
Arm/Group | Placebo | E6011 100 mg | E6011 200 mg | E6011 400/200 mg
Started | 56 | 29 | 54 | 55
Treated Participants | 54 | 28 | 54 | 54
Completed | 47 | 26 | 50 | 46
Not Completed | 9 | 3 | 4 | 9
Not completed — Inadequate Therapeutic Effect | 2 | 1 | 2 | 5
Not completed — Adverse Event | 2 | 1 | 0 | 3
Not completed — Progression of Disease | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Not Treated | 2 | 1 | 0 | 1
Period: Extension Phase (Open-label): 80 Weeks
Arm/Group | Placebo | E6011 100 mg | E6011 200 mg | E6011 400/200 mg
Started | 47 | 26 | 50 | 46
Completed | 36 | 17 | 36 | 35
Not Completed | 11 | 9 | 14 | 11
Not completed — Adverse Event | 1 | 2 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Inadequate Therapeutic Effect | 7 | 5 | 7 | 6
Not completed — Progression of Disease | 2 | 1 | 1 | 2
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement.
Groups:
- Placebo: During Treatment Phase, participants received E6011-matched placebo, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
- Total: Total of all reporting groups
Arm/Group | Placebo | E6011 100 mg | E6011 200 mg | E6011 400/200 mg | Total
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.86) | 56.5 (10.40) | 56.5 (10.39) | 55.2 (9.13) | 56.4 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 22 | 44 | 39 | 150
  Male | 9 | 6 | 10 | 15 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 28 | 54 | 54 | 190
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 54 | 28 | 54 | 54 | 190

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase: Percentage of Participants Who Achieved an American College of Rheumatology 20 (ACR20) Response at Week 12 Based on Non-responder Imputation (NRI)
Description: The ACR20 response was defined as if the following 3 criteria (ACR components) were met: Greater than or equal to (>=) 20 percent (%) reduction from baseline in the tender joint count (TJC) in 68 joints (TJC68); >=20% reduction from baseline in the swollen joint count (SJC) in 66 joints (SJC66); >=20% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (visual analog scale [VAS]) , Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), Health Assessment Questionnaire disability index (HAQ-DI), and C-reactive protein (CRP).
Time Frame: Week 12
Population: FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Missing data was imputed using NRI and this Outcome Measure was planned to be assessed only in Treatment Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment Phase: Placebo: During Treatment Phase, participants received E6011-matched placebo, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase.
- Treatment Phase: E6011 100 mg: During Treatment Phase, participants received E6011 100 mg, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase.
- Treatment Phase: E6011 200 mg: During Treatment Phase, participants received E6011 200 mg, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase.
- Treatment Phase: E6011 400/200 mg: During Treatment Phase, participants received E6011 400 mg, infusion, subcutaneously, at Weeks 0, 1, 4, 6, 8, 10 and then E6011 200 mg, infusion, subcutaneously, every 2 weeks up to Week 22. Following completion of evaluations of the Treatment Phase at Week 24, participants entered the Extension Phase.
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54
percentage of participants | 37.0 [24.16 to 49.92] | 39.3 [21.20 to 57.38] | 48.1 [34.82 to 61.47] | 46.3 [33.00 to 59.60]
Statistical Analysis 1: Comparison: Treatment Phase: Placebo vs Treatment Phase: E6011 100 mg; Test type: Superiority; p = 0.374, Regression, Logistic; Difference of arms = 2.2, 95% CI 2-sided [-19.96 to 24.46] — Estimate was calculated based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Treatment Phase: Placebo vs Treatment Phase: E6011 200 mg; Test type: Superiority; p = 0.102, Regression, Logistic; Difference of arms = 11.1, 95% CI 2-sided [-7.42 to 29.64] — Estimate was calculated based on the normal approximation to the binomial distribution
Statistical Analysis 3: Comparison: Treatment Phase: Placebo vs Treatment Phase: E6011 400/200 mg; Test type: Superiority; p = 0.188, Regression, Logistic; Difference of arms = 9.3, 95% CI 2-sided [-9.25 to 27.77] — Estimate was calculated based on the normal approximation to the binomial distribution

2. Secondary Outcome: Treatment Phase: Percentage of Participants Who Achieved an ACR20 Response at Weeks 2, 4, 8, 16, 20 and 24 Based on NRI
Description: The ACR20 response was defined as if the following 3 criteria (ACR components) were met: >=20% reduction from baseline in the TJC in 68 joints (TJC68); >=20% reduction from baseline in the SJC in 66 joints (SJC66); >=20% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (VAS), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), HAQ-DI, and CRP.
Time Frame: Weeks 2, 4, 8, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54
percentage of participants
  Response at Week 2 | 13.0 [4.00 to 21.92] | 14.3 [1.32 to 27.25] | 22.2 [11.13 to 33.31] | 20.4 [9.63 to 31.11]
  Response at Week 4 | 18.5 [8.16 to 28.88] | 28.6 [11.84 to 45.30] | 24.1 [12.67 to 35.48] | 31.5 [19.09 to 43.87]
  Response at Week 8 | 40.7 [27.64 to 53.85] | 35.7 [17.97 to 53.46] | 37.0 [24.16 to 49.92] | 46.3 [33.00 to 59.60]
  Response at Week 16 | 46.3 [33.00 to 59.60] | 46.4 [27.96 to 64.90] | 51.9 [38.53 to 65.18] | 53.7 [40.40 to 67.00]
  Response at Week 20 | 33.3 [20.76 to 45.91] | 50.0 [31.48 to 68.52] | 59.3 [46.15 to 72.36] | 55.6 [42.30 to 68.81]
  Response at Week 24 | 35.2 [22.45 to 47.92] | 39.3 [21.20 to 57.38] | 53.7 [40.40 to 67.00] | 57.4 [44.22 to 70.60]

3. Secondary Outcome: Treatment Phase: Percentage of Participants Who Achieved an ACR50 Response at Weeks 2, 4, 8, 16, 20 and 24 Based on NRI
Description: The ACR50 response was defined as if the following 3 criteria (ACR components) were met: >=50% reduction from baseline in the TJC in 68 joints (TJC68); >=50% reduction from baseline in the SJC in 66 joints (SJC66); >=50% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (VAS), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), HAQ-DI, and CRP.
Time Frame: Weeks 2, 4, 8, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54
percentage of participants
  Response at Week 2 | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 7.4 [0.42 to 14.39] | 7.4 [0.42 to 14.39]
  Response at Week 4 | 0.0 [0.00 to 0.00] | 3.6 [0.00 to 10.45] | 3.7 [0.00 to 8.74] | 9.3 [1.53 to 16.99]
  Response at Week 8 | 7.4 [0.42 to 14.39] | 14.3 [1.32 to 27.25] | 3.7 [0.00 to 8.74] | 9.3 [1.53 to 16.99]
  Response at Week 12 | 14.8 [5.34 to 24.29] | 10.7 [0.00 to 22.17] | 25.9 [14.24 to 37.61] | 18.5 [8.16 to 28.88]
  Response at Week 16 | 14.8 [5.34 to 24.29] | 17.9 [3.67 to 32.04] | 20.4 [9.63 to 31.11] | 22.2 [11.13 to 33.31]
  Response at Week 20 | 14.8 [5.34 to 24.29] | 10.7 [0.00 to 22.17] | 31.5 [19.09 to 43.87] | 25.9 [14.24 to 37.61]
  Response at Week 24 | 16.7 [6.73 to 26.61] | 17.9 [3.67 to 32.04] | 25.9 [14.24 to 37.61] | 27.8 [15.83 to 39.72]

4. Secondary Outcome: Treatment Phase: Percentage of Participants Who Achieved an ACR70 Response at Weeks 2, 4, 8, 16, 20 and 24 Based on NRI
Description: The ACR70 response was defined as if the following 3 criteria (ACR components) were met: >=70% reduction from baseline in the TJC in 68 joints (TJC68); >=70% reduction from baseline in the SJC in 66 joints (SJC66); >=70% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (VAS), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), HAQ-DI, and CRP.
Time Frame: Weeks 2, 4, 8, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54
percentage of participants
  Response at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00]
  Response at Week 4 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.9 [0.00 to 5.45]
  Response at Week 8 | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 5.6 [0.00 to 11.67]
  Response at Week 12 | 3.7 [0.00 to 8.74] | 3.6 [0.00 to 10.45] | 9.3 [1.53 to 16.99] | 7.4 [0.42 to 14.39]
  Response at Week 16 | 5.6 [0.00 to 11.67] | 7.1 [0.00 to 16.68] | 3.7 [0.00 to 8.74] | 13.0 [4.00 to 21.92]
  Response at Week 20 | 5.6 [0.00 to 11.67] | 7.1 [0.00 to 16.68] | 11.1 [2.73 to 19.49] | 14.8 [5.34 to 24.29]
  Response at Week 24 | 5.6 [0.00 to 11.67] | 14.3 [1.32 to 27.25] | 11.1 [2.73 to 19.49] | 13.0 [4.00 to 21.92]

5. Secondary Outcome: Change From Baseline in Tender Joint Counts (TJC) at Each Visit Based on Last Observation Carried Forward (LOCF)
Description: A total of 68 joints were examined for tenderness by applying pressure to the joint line or by moving joints through their respective ranges of motion. Joints were examined for tenderness by applying pressure to the joint line or by moving joints through their respective ranges of motion. Tender joints were marked with tick or cross in corresponding frames of the Assessment Sheet for Tender Joint Counts. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: Treatment Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24; Extension Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, and 84
Population: FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given time points. Missing data was imputed using LOCF imputation.
Measure: Mean (Standard Deviation); unit: tender joints
Groups:
- Extension Phase: Placebo: Participants who received E6011-matched placebo and completed evaluations of the Treatment Phase at Week 24, entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
- Extension Phase: E6011 100 mg: Participants who received E6011 100 mg and completed evaluations of the Treatment Phase at Week 24, entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
- Extension Phase: E6011 200 mg: Participants who received E6011 200 mg and completed evaluations of the Treatment Phase at Week 24, entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
- Extension Phase: E6011 400/200 mg: Participants who received E6011 400/200 mg and completed evaluations of the Treatment Phase at Week 24, entered the Extension Phase and received E6011 200 mg, infusion, subcutaneously, every 2 weeks until Week 102.
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
tender joints
  Baseline | 13.7 (6.81) | 14.1 (7.24) | 16.3 (7.15) | 16.6 (9.61) | 13.6 (6.72) | 14.3 (7.49) | 15.7 (6.70) | 16.6 (9.07)
  Change at Week 2 | -2.9 (5.63) | -2.7 (5.05) | -3.6 (5.99) | -3.9 (6.00) | -3.2 (4.88) | -2.5 (5.01) | -3.4 (5.99) | -4.5 (6.27)
  Change at Week 4 | -2.9 (6.04) | -2.9 (4.47) | -4.5 (5.34) | -5.8 (7.68) | -3.0 (5.63) | -2.8 (4.44) | -4.5 (5.29) | -6.7 (7.62)
  Change at Week 8 | -3.9 (7.00) | -4.6 (5.55) | -5.7 (6.14) | -6.7 (9.30) | -4.7 (6.12) | -4.6 (5.36) | -5.7 (5.98) | -7.6 (9.55)
  Change at Week 12 | -4.2 (7.40) | -5.2 (6.83) | -7.1 (7.42) | -7.9 (9.77) | -5.0 (6.54) | -5.3 (6.83) | -7.3 (7.18) | -8.9 (10.10)
  Change at Week 16 | -5.3 (7.51) | -6.4 (7.34) | -8.4 (6.53) | -7.9 (10.33) | -6.3 (6.53) | -6.6 (7.36) | -8.6 (6.20) | -9.3 (9.95)
  Change at Week 20 | -5.6 (8.50) | -6.9 (7.33) | -7.6 (7.72) | -8.5 (9.68) | -6.8 (7.70) | -7.2 (7.31) | -7.8 (7.59) | -10.0 (9.06)
  Change at Week 24 | -5.6 (7.97) | -6.9 (7.55) | -8.6 (7.38) | -8.7 (9.93) | -6.8 (7.02) | -7.2 (7.55) | -8.9 (7.13) | -10.4 (9.36)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -7.6 (7.85) | -7.5 (7.40) | -9.5 (7.74) | -10.1 (9.92)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -8.4 (7.94) | -7.9 (7.00) | -8.6 (7.94) | -10.0 (9.64)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -8.1 (9.25) | -7.6 (6.86) | -9.4 (6.85) | -11.3 (10.32)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -8.3 (8.98) | -7.5 (6.59) | -9.9 (6.79) | -10.7 (9.95)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -7.5 (8.12) | -7.4 (6.33) | -9.9 (7.53) | -11.4 (10.59)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -7.3 (9.30) | -8.2 (6.59) | -9.4 (7.98) | -10.9 (10.33)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -7.6 (7.90) | -8.0 (6.68) | -10.2 (6.44) | -10.7 (9.44)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -7.9 (7.65) | -7.7 (6.71) | -9.1 (7.62) | -11.0 (8.98)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -8.0 (8.03) | -8.4 (6.24) | -10.0 (8.14) | -11.5 (9.18)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -8.4 (8.70) | -8.7 (6.24) | -9.0 (7.86) | -12.1 (8.76)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -8.5 (8.15) | -7.5 (6.84) | -9.7 (8.45) | -12.0 (9.58)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -8.3 (8.23) | -7.9 (6.39) | -9.8 (7.80) | -11.2 (10.02)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -8.2 (8.12) | -8.2 (6.63) | -10.5 (7.88) | -11.8 (9.10)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -8.2 (8.29) | -8.5 (6.37) | -10.5 (7.77) | -11.8 (9.74)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -8.2 (8.08) | -8.0 (6.26) | -10.5 (7.79) | -11.7 (9.99)

6. Secondary Outcome: Change From Baseline in Swollen Joint Counts (SJC) at Each Visit Based on LOCF
Description: A total of 66 joints (minus 2 hip joints from evaluated tender joints) were examined for swollen joints. Swollen joints were marked with open circles in corresponding frames of the Assessment Sheet for Swollen Joint Counts. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
swollen joints
  Baseline | 12.7 (6.81) | 11.3 (5.27) | 12.4 (4.89) | 13.5 (6.41) | 12.7 (6.48) | 11.5 (5.38) | 12.1 (4.63) | 13.8 (6.18)
  Change at Week 2 | -2.2 (4.70) | -2.8 (3.33) | -2.9 (4.18) | -3.4 (5.25) | -2.9 (4.21) | -2.9 (3.46) | -3.0 (3.84) | -3.7 (5.17)
  Change at Week 4 | -3.0 (5.36) | -3.7 (3.42) | -3.3 (4.66) | -5.0 (4.95) | -3.8 (3.94) | -3.8 (3.51) | -3.5 (4.03) | -5.5 (5.01)
  Change at Week 8 | -4.1 (7.33) | -4.7 (4.16) | -3.8 (5.82) | -6.0 (5.81) | -5.7 (4.70) | -4.7 (4.32) | -3.8 (5.42) | -6.7 (5.74)
  Change at Week 12 | -4.2 (7.05) | -5.1 (4.91) | -4.9 (5.39) | -5.7 (6.41) | -5.9 (4.11) | -5.2 (5.08) | -5.2 (4.93) | -6.4 (6.34)
  Change at Week 16 | -4.3 (7.38) | -6.1 (4.32) | -5.2 (5.30) | -6.6 (6.60) | -6.0 (4.65) | -6.3 (4.43) | -5.5 (4.81) | -8.0 (5.68)
  Change at Week 20 | -5.1 (8.73) | -6.4 (4.65) | -5.6 (5.71) | -6.4 (7.26) | -7.0 (6.50) | -6.6 (4.78) | -5.8 (5.28) | -7.7 (6.61)
  Change at Week 24 | -5.1 (8.32) | -6.3 (4.28) | -5.9 (6.38) | -6.2 (6.65) | -7.0 (5.86) | -6.5 (4.38) | -6.2 (5.93) | -7.6 (5.74)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -7.2 (6.77) | -7.8 (5.05) | -6.9 (5.71) | -8.5 (5.98)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -7.9 (7.04) | -7.6 (4.63) | -7.0 (6.17) | -8.6 (6.31)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -7.2 (7.52) | -7.5 (4.64) | -7.1 (5.90) | -9.0 (5.75)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -7.4 (7.55) | -7.2 (4.43) | -6.8 (5.10) | -8.4 (5.64)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -6.9 (7.75) | -6.5 (4.54) | -6.8 (5.44) | -8.3 (6.32)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -7.2 (8.04) | -6.7 (4.48) | -6.4 (6.11) | -8.5 (5.82)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -7.2 (7.19) | -6.7 (4.54) | -6.3 (5.03) | -8.3 (5.30)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -7.3 (7.18) | -7.0 (3.77) | -6.3 (5.89) | -8.6 (5.70)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -7.4 (6.83) | -7.3 (4.32) | -6.5 (6.40) | -8.5 (6.17)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -7.5 (7.67) | -7.3 (4.61) | -6.4 (6.21) | -8.5 (5.75)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -8.0 (7.30) | -6.5 (5.21) | -6.9 (5.79) | -8.6 (5.78)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -7.9 (7.49) | -7.0 (4.76) | -6.9 (5.93) | -8.8 (5.68)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -7.7 (7.21) | -6.3 (4.77) | -7.1 (5.81) | -8.3 (5.59)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -7.2 (7.50) | -7.1 (4.89) | -6.7 (6.18) | -8.4 (6.07)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -7.7 (7.38) | -7.2 (4.92) | -6.9 (6.08) | -8.2 (6.25)

7. Secondary Outcome: Change From Baseline in Participant's Assessment of Pain Based on VAS Score at Each Visit Based on LOCF
Description: Intensity and severity of pain associated with rheumatoid arthritis (RA) were indicated by the participant on a score sheet, Pain/disease activity assessments reported by the participant, by placing a mark on a 100 millimeter (mm) horizontal VAS. The scale ranged from 0-100 mm, where 0 indicated no disease activity (symptom free and no arthritis symptoms) and 100 represented maximum disease activity (maximum arthritis disease activity). Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
units on a scale
  Baseline | 53.6 (23.03) | 47.9 (26.37) | 46.6 (23.03) | 52.9 (24.38) | 54.2 (21.89) | 46.6 (26.94) | 46.7 (22.95) | 49.6 (24.25)
  Change at Week 2 | -4.0 (17.96) | -4.5 (12.64) | -6.2 (17.22) | -5.9 (16.91) | -5.2 (18.88) | -4.4 (13.08) | -6.4 (17.81) | -5.1 (17.00)
  Change at Week 4 | -5.8 (22.47) | -6.4 (20.68) | -4.1 (18.36) | -9.0 (18.93) | -9.0 (21.34) | -6.6 (21.47) | -4.4 (18.77) | -8.3 (19.19)
  Change at Week 8 | -7.8 (20.76) | -4.9 (19.96) | -10.0 (18.29) | -16.6 (22.58) | -10.5 (18.73) | -5.7 (20.51) | -11.0 (18.45) | -17.0 (23.50)
  Change at Week 12 | -7.5 (26.09) | -12.2 (18.19) | -12.9 (21.24) | -13.7 (25.24) | -11.0 (25.10) | -12.8 (18.75) | -14.6 (20.72) | -15.2 (26.57)
  Change at Week 16 | -10.8 (27.25) | -11.4 (19.69) | -13.6 (20.87) | -15.1 (25.78) | -14.1 (26.26) | -11.7 (20.42) | -14.8 (20.91) | -17.8 (26.62)
  Change at Week 20 | -9.1 (29.43) | -13.5 (19.33) | -15.0 (21.08) | -16.6 (26.04) | -12.9 (28.35) | -14.4 (19.75) | -16.6 (20.67) | -19.3 (26.67)
  Change at Week 24 | -9.4 (28.49) | -13.9 (21.59) | -14.4 (20.85) | -18.5 (24.29) | -13.2 (27.17) | -14.8 (22.11) | -16.0 (20.47) | -21.6 (24.35)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -18.0 (26.34) | -12.9 (25.13) | -14.0 (22.45) | -22.3 (27.16)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -17.9 (27.27) | -16.9 (23.06) | -14.6 (22.57) | -21.0 (33.28)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -15.5 (28.89) | -14.4 (23.58) | -16.8 (25.04) | -22.2 (31.15)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -15.3 (28.08) | -15.5 (23.14) | -17.7 (23.93) | -22.7 (29.17)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -16.7 (26.93) | -17.8 (21.77) | -17.5 (23.27) | -23.1 (29.58)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -20.0 (27.74) | -17.6 (24.36) | -17.6 (22.50) | -23.4 (28.36)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -17.2 (28.24) | -15.3 (25.63) | -16.9 (25.39) | -22.7 (24.17)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -20.8 (27.88) | -16.0 (25.02) | -18.7 (22.74) | -21.8 (24.98)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -22.6 (28.21) | -16.2 (23.69) | -18.0 (23.76) | -24.6 (26.90)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -21.2 (26.46) | -16.1 (24.34) | -17.5 (26.63) | -22.0 (26.80)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -24.6 (27.59) | -17.7 (25.96) | -16.2 (25.65) | -24.1 (27.79)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -23.3 (27.81) | -16.7 (24.96) | -16.2 (25.49) | -24.5 (27.82)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -21.4 (27.70) | -19.0 (26.29) | -16.9 (25.92) | -24.2 (28.00)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -21.4 (29.20) | -19.3 (25.29) | -16.2 (25.09) | -24.8 (25.53)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -23.2 (28.58) | -18.3 (26.01) | -17.1 (24.50) | -24.4 (27.29)

8. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity Based on VAS Score at Each Visit Based on LOCF
Description: Participants were evaluated on their disease activity of RA, and entered the result on the score sheet, disease activity assessments reported by the participant, by placing a mark on a 100 mm horizontal VAS. The scale ranged from 0-100 mm, where 0 indicated no disease activity (symptom free and no arthritis symptoms) and 100 represented maximum disease activity (maximum arthritis disease activity). Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
units on a scale
  Baseline | 53.1 (25.74) | 50.1 (25.04) | 49.0 (22.37) | 54.5 (23.97) | 53.4 (25.30) | 49.2 (25.77) | 49.2 (22.19) | 51.3 (23.89)
  Change at Week 2 | -2.9 (20.03) | -4.2 (14.32) | -8.3 (17.32) | -6.4 (16.40) | -3.8 (21.28) | -4.5 (14.70) | -8.5 (17.84) | -5.5 (16.45)
  Change at Week 4 | -6.4 (24.49) | -6.6 (17.03) | -7.2 (16.29) | -9.8 (19.73) | -9.4 (23.96) | -7.0 (17.50) | -7.6 (16.64) | -9.5 (20.26)
  Change at Week 8 | -5.5 (23.48) | -7.3 (18.62) | -11.6 (18.67) | -18.1 (23.66) | -7.5 (22.61) | -8.5 (18.82) | -12.8 (18.80) | -18.8 (24.76)
  Change at Week 12 | -7.3 (27.83) | -14.6 (18.22) | -15.2 (18.50) | -15.1 (27.23) | -10.0 (27.59) | -15.8 (18.36) | -17.0 (17.62) | -17.3 (28.74)
  Change at Week 16 | -11.6 (27.40) | -14.0 (20.19) | -16.1 (20.49) | -16.6 (27.22) | -14.7 (26.47) | -15.3 (20.31) | -17.4 (20.46) | -19.3 (28.40)
  Change at Week 20 | -10.0 (30.67) | -15.3 (19.24) | -17.4 (21.43) | -17.8 (28.14) | -13.6 (29.69) | -17.0 (18.89) | -19.2 (21.03) | -20.7 (29.30)
  Change at Week 24 | -8.8 (30.97) | -15.3 (23.29) | -17.8 (20.27) | -20.4 (24.90) | -12.3 (30.20) | -17.0 (23.30) | -19.6 (19.72) | -23.8 (25.11)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -17.1 (30.18) | -17.0 (24.50) | -18.5 (21.28) | -24.8 (27.56)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -19.3 (29.27) | -19.8 (20.81) | -16.7 (24.64) | -23.2 (32.64)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -15.7 (28.40) | -17.0 (22.63) | -19.6 (24.05) | -24.2 (31.25)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -15.8 (30.76) | -18.6 (21.01) | -20.4 (23.40) | -24.6 (29.17)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -16.9 (27.20) | -20.3 (20.23) | -20.2 (23.05) | -25.0 (29.55)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -18.5 (28.84) | -19.6 (22.90) | -20.3 (20.80) | -24.8 (29.19)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -16.1 (31.20) | -17.0 (23.15) | -19.4 (23.97) | -24.6 (25.27)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -20.0 (29.52) | -18.0 (23.09) | -20.3 (21.95) | -25.2 (27.24)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -21.3 (28.76) | -19.0 (21.14) | -20.8 (23.05) | -26.3 (27.92)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -20.1 (27.01) | -19.1 (23.63) | -19.9 (24.04) | -24.5 (27.89)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -22.9 (28.89) | -19.5 (25.09) | -18.6 (24.69) | -26.9 (28.56)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -21.7 (31.19) | -19.0 (24.98) | -18.6 (25.14) | -26.4 (28.61)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -21.3 (29.79) | -20.9 (24.88) | -20.3 (25.11) | -26.2 (28.19)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -21.0 (30.98) | -20.4 (24.23) | -19.2 (23.56) | -27.3 (27.01)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -21.1 (31.62) | -19.6 (24.67) | -19.6 (22.45) | -27.0 (28.96)

9. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity Scale Based on VAS Score at Each Visit Based on LOCF
Description: The Physician's Global Assessment of Disease Activity was recorded using the 100 mm horizontal VAS. Physician rated participant's RA disease activity on a scale ranged from 0-100 mm, where 0 indicated no disease activity (no arthritis) and 100 represented maximum disease activity (maximum arthritis). Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
units on a scale
  Baseline | 54.3 (19.07) | 53.1 (21.88) | 55.2 (17.27) | 54.2 (22.02) | 53.7 (19.17) | 52.0 (22.20) | 54.2 (17.30) | 53.9 (21.28)
  Change at Week 2 | -10.1 (15.95) | -9.5 (16.32) | -11.1 (15.59) | -7.9 (16.61) | -10.4 (14.73) | -7.3 (14.59) | -10.3 (15.78) | -8.1 (17.63)
  Change at Week 4 | -8.4 (16.83) | -7.6 (14.11) | -15.2 (16.36) | -13.2 (20.76) | -9.9 (15.99) | -6.7 (13.23) | -15.0 (16.68) | -13.8 (21.74)
  Change at Week 8 | -13.6 (21.08) | -11.3 (16.87) | -16.6 (20.75) | -16.1 (21.51) | -15.5 (17.70) | -9.3 (15.25) | -16.7 (21.00) | -19.0 (21.63)
  Change at Week 12 | -14.9 (24.14) | -16.9 (24.74) | -21.6 (18.54) | -18.1 (26.27) | -17.1 (21.36) | -16.8 (25.04) | -22.3 (17.53) | -19.5 (26.63)
  Change at Week 16 | -16.1 (23.49) | -19.3 (20.88) | -23.1 (20.21) | -19.3 (25.83) | -19.1 (21.49) | -19.3 (20.91) | -23.6 (20.00) | -23.7 (23.80)
  Change at Week 20 | -15.3 (25.97) | -20.0 (21.27) | -22.7 (20.32) | -18.9 (28.39) | -18.8 (24.20) | -20.9 (21.65) | -23.3 (19.81) | -23.1 (27.08)
  Change at Week 24 | -15.5 (26.23) | -17.8 (24.33) | -24.6 (21.38) | -20.8 (27.39) | -19.0 (24.49) | -18.4 (24.96) | -25.4 (20.91) | -25.7 (25.19)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -24.4 (22.28) | -20.1 (24.68) | -28.1 (19.69) | -27.4 (26.36)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -25.9 (25.28) | -21.7 (26.24) | -24.4 (21.13) | -25.9 (26.01)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -23.9 (25.96) | -19.3 (23.02) | -25.3 (20.46) | -29.2 (27.19)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -25.2 (26.39) | -22.7 (25.52) | -27.8 (16.77) | -27.0 (27.64)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -25.8 (28.22) | -19.8 (22.76) | -27.6 (19.34) | -29.2 (28.51)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -27.3 (29.35) | -21.6 (25.58) | -27.8 (20.44) | -26.9 (29.34)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -23.3 (28.22) | -19.9 (24.81) | -26.7 (20.55) | -26.8 (28.30)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -23.6 (25.87) | -20.8 (24.91) | -26.8 (19.72) | -28.2 (26.27)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -23.9 (28.72) | -21.1 (23.93) | -27.0 (21.24) | -29.7 (26.70)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -26.4 (28.15) | -20.1 (22.32) | -24.9 (21.16) | -29.4 (25.93)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -27.9 (27.73) | -21.6 (26.92) | -27.4 (21.10) | -30.3 (27.03)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -25.0 (28.10) | -20.2 (22.55) | -27.1 (22.45) | -29.0 (25.74)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -23.5 (28.17) | -22.4 (22.89) | -27.6 (21.89) | -31.2 (26.22)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -24.0 (28.33) | -24.9 (26.05) | -26.9 (21.29) | -31.5 (25.95)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -25.9 (28.47) | -21.8 (24.09) | -27.3 (20.49) | -30.1 (25.70)

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Each Visit Based on LOCF
Description: The degree of disability was self-evaluated by the participant using the HAQ-DI. The assessment was made based on the activities capable without any aids or devices. The 20-question instrument assessed the degree of difficulty a person had in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0, indicated no difficulty, to 3, indicated inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range: 0-3 where 0 = least difficulty and 3 = extreme difficulty. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
units on a scale
  Baseline | 0.77 (0.526) | 0.73 (0.527) | 0.75 (0.602) | 0.80 (0.611) | 0.75 (0.519) | 0.72 (0.541) | 0.74 (0.618) | 0.71 (0.543)
  Change at Week 2 | 0.00 (0.281) | -0.01 (0.236) | -0.06 (0.295) | -0.06 (0.301) | -0.03 (0.223) | 0.00 (0.240) | -0.05 (0.297) | -0.05 (0.306)
  Change at Week 4 | 0.02 (0.352) | 0.01 (0.277) | -0.07 (0.299) | -0.10 (0.303) | -0.02 (0.265) | 0.03 (0.281) | -0.06 (0.301) | -0.12 (0.304)
  Change at Week 8 | 0.00 (0.432) | -0.03 (0.298) | -0.10 (0.323) | -0.12 (0.329) | -0.03 (0.379) | -0.03 (0.296) | -0.08 (0.319) | -0.13 (0.350)
  Change at Week 12 | 0.01 (0.493) | -0.06 (0.356) | -0.13 (0.321) | -0.14 (0.402) | -0.02 (0.463) | -0.04 (0.351) | -0.11 (0.321) | -0.16 (0.422)
  Change at Week 16 | -0.03 (0.469) | -0.08 (0.330) | -0.19 (0.330) | -0.13 (0.411) | -0.06 (0.434) | -0.06 (0.315) | -0.18 (0.332) | -0.15 (0.433)
  Change at Week 20 | 0.02 (0.519) | -0.10 (0.285) | -0.17 (0.335) | -0.14 (0.435) | -0.03 (0.485) | -0.09 (0.285) | -0.17 (0.337) | -0.16 (0.461)
  Change at Week 24 | -0.02 (0.494) | -0.09 (0.300) | -0.17 (0.337) | -0.17 (0.446) | -0.07 (0.450) | -0.08 (0.300) | -0.16 (0.339) | -0.20 (0.470)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -0.07 (0.523) | -0.09 (0.278) | -0.21 (0.407) | -0.23 (0.479)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -0.11 (0.544) | -0.13 (0.314) | -0.18 (0.392) | -0.10 (0.670)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -0.05 (0.547) | -0.06 (0.396) | -0.20 (0.381) | -0.17 (0.614)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -0.05 (0.531) | -0.08 (0.337) | -0.17 (0.318) | -0.19 (0.594)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -0.10 (0.544) | -0.11 (0.380) | -0.19 (0.415) | -0.19 (0.561)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -0.08 (0.546) | -0.06 (0.366) | -0.20 (0.434) | -0.20 (0.592)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -0.06 (0.535) | -0.04 (0.318) | -0.22 (0.385) | -0.19 (0.549)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -0.09 (0.525) | -0.06 (0.303) | -0.20 (0.425) | -0.20 (0.539)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -0.10 (0.551) | -0.09 (0.297) | -0.19 (0.422) | -0.24 (0.567)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -0.09 (0.518) | -0.06 (0.366) | -0.13 (0.457) | -0.25 (0.591)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -0.13 (0.559) | -0.09 (0.356) | -0.16 (0.508) | -0.24 (0.597)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -0.17 (0.542) | -0.06 (0.357) | -0.19 (0.500) | -0.23 (0.596)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -0.16 (0.557) | -0.11 (0.309) | -0.18 (0.475) | -0.26 (0.602)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -0.11 (0.555) | -0.12 (0.325) | -0.16 (0.514) | -0.25 (0.579)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -0.15 (0.567) | -0.08 (0.332) | -0.19 (0.467) | -0.25 (0.586)

11. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Values at Each Visit Based on LOCF
Description: CRP of each participants was measured as a part of blood biochemical tests. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
milligram per deciliter (mg/dL)
  Baseline | 1.50 (1.633) | 1.44 (1.868) | 1.08 (0.840) | 1.24 (1.634) | 1.42 (1.682) | 1.41 (1.901) | 1.04 (0.843) | 1.07 (1.291)
  Change at Week 2 | -0.09 (0.909) | -0.28 (1.148) | 0.08 (0.707) | 0.07 (0.777) | -0.16 (0.930) | -0.32 (1.176) | 0.08 (0.715) | 0.12 (0.769)
  Change at Week 4 | 0.06 (1.235) | 0.20 (1.279) | 0.04 (0.707) | 0.33 (1.383) | -0.14 (1.134) | 0.15 (1.268) | 0.03 (0.694) | 0.28 (1.443)
  Change at Week 8 | 0.21 (1.192) | 0.12 (1.750) | 0.29 (1.407) | -0.03 (1.343) | 0.04 (1.103) | 0.08 (1.787) | 0.28 (1.452) | -0.15 (1.392)
  Change at Week 12 | 0.15 (1.503) | -0.23 (1.429) | -0.06 (1.263) | -0.05 (1.403) | 0.01 (1.485) | -0.26 (1.481) | -0.07 (1.309) | -0.24 (1.314)
  Change at Week 16 | 0.17 (1.429) | -0.26 (1.626) | -0.11 (1.214) | 0.09 (1.737) | 0.00 (1.412) | -0.29 (1.684) | -0.10 (1.249) | -0.08 (1.713)
  Change at Week 20 | 0.24 (1.686) | -0.17 (1.683) | -0.18 (1.071) | 0.01 (1.332) | 0.00 (1.652) | -0.25 (1.712) | -0.23 (1.060) | -0.14 (1.154)
  Change at Week 24 | 0.39 (2.063) | -0.26 (1.887) | 0.01 (1.155) | 0.38 (2.220) | 0.18 (2.106) | -0.35 (1.924) | -0.03 (1.161) | 0.30 (2.269)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -0.24 (1.792) | -0.34 (1.603) | -0.21 (0.997) | -0.19 (1.677)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -0.10 (2.067) | -0.32 (1.617) | 0.13 (1.585) | -0.35 (1.371)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -0.10 (1.839) | -0.13 (2.311) | -0.04 (1.301) | -0.24 (1.691)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -0.17 (1.852) | -0.30 (1.801) | -0.10 (1.100) | -0.25 (1.539)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -0.10 (1.939) | -0.35 (1.908) | 0.26 (1.798) | -0.17 (1.470)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | 0.14 (1.910) | -0.25 (2.131) | -0.04 (1.103) | -0.32 (1.416)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | 0.33 (2.130) | -0.23 (2.288) | -0.10 (1.134) | -0.14 (1.162)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -0.09 (1.967) | -0.44 (2.001) | -0.03 (1.264) | -0.27 (1.124)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -0.13 (1.956) | -0.14 (2.375) | -0.03 (1.266) | -0.39 (1.276)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -0.04 (2.062) | -0.34 (2.115) | 0.54 (4.066) | -0.40 (1.307)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -0.26 (2.207) | -0.23 (2.276) | 0.13 (1.662) | -0.36 (1.414)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -0.17 (2.414) | -0.27 (2.167) | 0.04 (1.550) | -0.28 (1.437)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -0.09 (2.382) | -0.38 (2.115) | 0.07 (1.593) | -0.41 (1.329)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -0.20 (2.297) | -0.32 (2.065) | 0.02 (1.524) | -0.40 (1.260)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -0.23 (2.332) | -0.39 (2.097) | 0.11 (1.754) | -0.35 (1.417)

12. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) Values at Each Visit Based on LOCF
Description: ESR were a type of blood test. An ESR was used to monitor the arthritis condition. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: Treatment Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24; Extension Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80,and 84
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter per hour (mm/hr)
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
millimeter per hour (mm/hr)
  Baseline | 41.6 (26.37) | 37.9 (16.62) | 40.8 (20.06) | 40.1 (20.45) | 39.6 (26.47) | 37.6 (17.21) | 40.0 (19.67) | 38.3 (16.91)
  Change at Week 2 | -3.8 (10.40) | 1.0 (8.25) | -1.9 (7.53) | 0.7 (10.38) | -4.1 (10.49) | 1.7 (8.00) | -2.1 (7.70) | 0.4 (10.92)
  Change at Week 4 | -2.3 (14.51) | 1.3 (11.79) | -2.6 (7.42) | -1.1 (13.38) | -3.4 (14.07) | 1.3 (12.22) | -2.8 (7.62) | -2.2 (13.49)
  Change at Week 8 | 0.2 (17.72) | -0.3 (11.62) | -1.8 (14.43) | -3.7 (15.09) | -1.5 (16.90) | -0.5 (11.55) | -2.7 (14.19) | -5.3 (15.29)
  Change at Week 12 | -0.3 (16.46) | -2.9 (15.53) | -3.8 (18.39) | -3.5 (17.83) | -1.5 (15.28) | -3.4 (16.00) | -4.7 (18.38) | -5.7 (17.77)
  Change at Week 16 | -1.9 (15.78) | -3.3 (18.53) | -5.5 (20.68) | -2.2 (19.92) | -3.6 (14.47) | -3.8 (19.14) | -6.0 (21.05) | -4.7 (20.03)
  Change at Week 20 | -0.6 (22.08) | -1.3 (18.75) | -6.6 (20.32) | -4.0 (19.17) | -2.3 (21.23) | -2.3 (19.00) | -8.0 (19.80) | -6.8 (18.86)
  Change at Week 24 | -0.1 (23.16) | 0.6 (20.14) | -4.0 (21.67) | -2.9 (20.41) | -1.8 (22.56) | -0.3 (20.57) | -5.2 (21.47) | -5.4 (20.52)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -4.6 (20.04) | -4.3 (19.51) | -3.4 (23.67) | -8.0 (18.76)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -3.4 (21.50) | -5.0 (16.34) | -3.9 (23.50) | -7.4 (20.18)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -4.7 (20.43) | -4.5 (20.44) | -1.9 (23.56) | -4.8 (20.81)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -3.4 (19.46) | -3.5 (19.77) | -3.1 (24.00) | -5.8 (21.58)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -3.2 (20.19) | -4.4 (21.73) | -3.2 (24.65) | -4.8 (22.59)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -2.0 (19.12) | -2.0 (20.91) | -4.2 (20.41) | -5.5 (19.42)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -0.6 (19.64) | -1.8 (21.69) | -2.5 (25.04) | -4.9 (20.18)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -4.6 (21.59) | -4.4 (20.37) | -3.9 (23.46) | -6.2 (19.83)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -4.9 (22.00) | -2.6 (23.13) | -3.6 (26.27) | -7.6 (19.37)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -4.1 (24.32) | -3.2 (22.29) | -5.5 (24.06) | -8.0 (18.98)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -4.0 (24.77) | -3.2 (22.21) | -5.9 (22.68) | -8.7 (17.98)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -4.5 (27.08) | -3.7 (20.94) | -4.3 (24.37) | -7.8 (20.01)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -4.2 (26.28) | -4.8 (18.96) | -4.4 (22.94) | -7.9 (18.92)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -5.7 (27.22) | -4.6 (19.36) | -6.1 (24.45) | -9.1 (18.06)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -5.9 (25.74) | -5.1 (19.08) | -3.0 (24.74) | -8.1 (18.95)

13. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28)-ESR Values at Each Visit Based on LOCF
Description: The DAS28 index was a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and ESR value. Total score ranged between 0-10. A DAS28-ESR score of 5.1 or above = high disease activity, a value between 3.2 and 5.1 = moderate disease activity and value between 2.6 and 3.2 = low disease activity, value <2.6 = disease remission. A positive change in score indicates worsening, and a negative change indicates improvement. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
score on a scale
  Baseline | 5.709 (0.9161) | 5.687 (0.9278) | 5.819 (0.7696) | 5.984 (0.8865) | 5.653 (0.9149) | 5.674 (0.9625) | 5.775 (0.6980) | 5.931 (0.8490)
  Change at Week 2 | -0.520 (0.7531) | -0.402 (0.5058) | -0.554 (0.6165) | -0.420 (0.6906) | -0.580 (0.7398) | -0.392 (0.4917) | -0.541 (0.6199) | -0.436 (0.7121)
  Change at Week 4 | -0.571 (0.8416) | -0.434 (0.6825) | -0.702 (0.6534) | -0.833 (1.0092) | -0.641 (0.8217) | -0.423 (0.6709) | -0.710 (0.6435) | -0.896 (1.0426)
  Change at Week 8 | -0.674 (1.1682) | -0.642 (0.8081) | -0.919 (0.8813) | -1.217 (1.1963) | -0.839 (1.0703) | -0.653 (0.7871) | -0.947 (0.8681) | -1.306 (1.2425)
  Change at Week 12 | -0.763 (1.2561) | -1.007 (1.0644) | -1.237 (1.0536) | -1.277 (1.4323) | -0.934 (1.1527) | -1.053 (1.0693) | -1.302 (0.9895) | -1.443 (1.4777)
  Change at Week 16 | -1.022 (1.3026) | -1.134 (1.1573) | -1.391 (1.0674) | -1.349 (1.4847) | -1.242 (1.1588) | -1.195 (1.1625) | -1.445 (1.0294) | -1.581 (1.4581)
  Change at Week 20 | -0.977 (1.3914) | -1.156 (1.0949) | -1.449 (1.2393) | -1.525 (1.4998) | -1.215 (1.2400) | -1.226 (1.0921) | -1.524 (1.1984) | -1.787 (1.4405)
  Change at Week 24 | -0.950 (1.4587) | -1.144 (1.2704) | -1.470 (1.1853) | -1.536 (1.5340) | -1.185 (1.3317) | -1.214 (1.2817) | -1.546 (1.1363) | -1.815 (1.4668)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -1.452 (1.3306) | -1.397 (1.3890) | -1.652 (1.2452) | -1.913 (1.4510)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -1.512 (1.3217) | -1.457 (1.2777) | -1.617 (1.4220) | -1.856 (1.5063)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -1.443 (1.3900) | -1.336 (1.3160) | -1.718 (1.2962) | -1.994 (1.5330)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -1.409 (1.3896) | -1.362 (1.3332) | -1.672 (1.1859) | -1.947 (1.5247)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -1.367 (1.3085) | -1.391 (1.2689) | -1.727 (1.2501) | -2.063 (1.5432)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -1.438 (1.4786) | -1.447 (1.3270) | -1.734 (1.2812) | -2.004 (1.4325)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -1.387 (1.4577) | -1.364 (1.2433) | -1.682 (1.1280) | -1.956 (1.4547)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -1.516 (1.4242) | -1.398 (1.2493) | -1.678 (1.2286) | -2.122 (1.4580)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -1.528 (1.4876) | -1.579 (1.3403) | -1.764 (1.4278) | -2.145 (1.4990)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -1.483 (1.4218) | -1.538 (1.2862) | -1.652 (1.3363) | -2.188 (1.4525)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -1.598 (1.4828) | -1.411 (1.3355) | -1.729 (1.4047) | -2.221 (1.4155)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -1.528 (1.5740) | -1.402 (1.2321) | -1.742 (1.3978) | -2.100 (1.4930)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -1.547 (1.6002) | -1.458 (1.1877) | -1.833 (1.3346) | -2.133 (1.3671)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -1.580 (1.6735) | -1.544 (1.2228) | -1.773 (1.2908) | -2.194 (1.4738)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -1.599 (1.5656) | -1.584 (1.3414) | -1.812 (1.3174) | -2.206 (1.5263)

14. Secondary Outcome: Change From Baseline in DAS28-CRP Values at Each Visit Based on LOCF
Description: The DAS28 index was a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and CRP value. Total score ranged between 0-10. A DAS28-CRP score of 5.1 or above = high disease activity, a value between 3.2 and 5.1 = moderate disease activity and value between 2.6 and 3.2 = low disease activity, value <2.6 = disease remission. A positive change in score indicates worsening, and a negative change indicates improvement. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
score on a scale
  Baseline | 5.039 (0.8789) | 4.993 (1.0096) | 5.079 (0.7290) | 5.202 (0.9283) | 4.997 (0.8561) | 4.978 (1.0458) | 5.034 (0.6676) | 5.138 (0.8998)
  Change at Week 2 | -0.474 (0.7500) | -0.464 (0.5214) | -0.531 (0.6404) | -0.430 (0.7393) | -0.534 (0.7370) | -0.459 (0.5043) | -0.514 (0.6403) | -0.433 (0.7731)
  Change at Week 4 | -0.514 (0.8858) | -0.407 (0.6521) | -0.675 (0.6705) | -0.704 (0.9959) | -0.591 (0.8735) | -0.391 (0.6202) | -0.678 (0.6539) | -0.747 (1.0501)
  Change at Week 8 | -0.607 (1.0640) | -0.679 (0.8212) | -0.885 (0.8535) | -1.059 (1.1604) | -0.767 (0.9529) | -0.684 (0.7985) | -0.905 (0.8341) | -1.136 (1.2236)
  Change at Week 12 | -0.692 (1.2057) | -1.028 (1.0399) | -1.206 (1.0564) | -1.164 (1.3302) | -0.855 (1.0981) | -1.071 (1.0433) | -1.260 (1.0062) | -1.321 (1.3768)
  Change at Week 16 | -0.913 (1.2429) | -1.160 (1.0453) | -1.339 (1.0190) | -1.250 (1.4208) | -1.125 (1.1056) | -1.222 (1.0420) | -1.385 (0.9817) | -1.473 (1.3859)
  Change at Week 20 | -0.889 (1.3450) | -1.186 (1.0136) | -1.397 (1.2380) | -1.437 (1.4440) | -1.133 (1.1959) | -1.264 (1.0004) | -1.461 (1.2066) | -1.692 (1.3754)
  Change at Week 24 | -0.825 (1.3502) | -1.212 (1.1955) | -1.449 (1.1679) | -1.400 (1.4462) | -1.058 (1.2175) | -1.292 (1.1959) | -1.518 (1.1251) | -1.666 (1.3715)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -1.363 (1.2248) | -1.386 (1.2327) | -1.645 (1.2490) | -1.770 (1.3779)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -1.438 (1.2821) | -1.461 (1.1617) | -1.545 (1.4075) | -1.724 (1.4062)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -1.319 (1.2935) | -1.329 (1.2331) | -1.729 (1.2139) | -1.910 (1.4317)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -1.343 (1.3170) | -1.359 (1.1999) | -1.688 (1.0828) | -1.835 (1.4415)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -1.286 (1.2637) | -1.334 (1.1039) | -1.702 (1.2073) | -1.915 (1.5062)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -1.338 (1.4080) | -1.475 (1.2492) | -1.658 (1.1945) | -1.904 (1.3723)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -1.293 (1.4043) | -1.407 (1.1550) | -1.660 (1.1057) | -1.815 (1.2919)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -1.425 (1.3826) | -1.438 (1.1264) | -1.603 (1.2139) | -1.999 (1.3047)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -1.392 (1.4082) | -1.557 (1.1507) | -1.697 (1.3250) | -2.015 (1.3216)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -1.380 (1.3475) | -1.530 (1.1474) | -1.579 (1.2837) | -2.039 (1.2069)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -1.520 (1.4072) | -1.414 (1.2456) | -1.627 (1.3523) | -2.092 (1.2697)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -1.434 (1.4852) | -1.398 (1.1240) | -1.698 (1.2813) | -1.946 (1.3801)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -1.445 (1.5266) | -1.489 (1.1022) | -1.783 (1.2366) | -2.029 (1.2583)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -1.438 (1.5290) | -1.544 (1.1475) | -1.688 (1.1779) | -2.069 (1.3821)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -1.524 (1.5688) | -1.596 (1.2642) | -1.750 (1.2376) | -2.090 (1.4318)

15. Secondary Outcome: Change From Baseline in Simple Disease Activity Index (SDAI) Values at Each Visit Based on LOCF
Description: The SDAI was calculated from tender joint counts of 28, swollen joint counts of 28, participant's global assessment of disease activity, physician global assessment of disease activity score, and CRP value. Total score ranged between 0-86. SDAI score of 26 or above = high disease activity, a value between 11 and 26 = moderate disease activity and value less than or equal to (<=) 11 = low disease activity, value <=33 = disease remission. Higher scores indicated higher disease activity. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
score on a scale
  Baseline | 30.694 (10.7598) | 30.546 (12.5152) | 31.646 (9.3821) | 34.413 (12.6292) | 30.317 (10.5425) | 30.604 (12.9983) | 30.962 (8.2366) | 33.915 (11.9378)
  Change at Week 2 | -5.093 (8.0941) | -5.618 (6.0585) | -6.704 (6.9970) | -6.352 (9.5528) | -5.800 (6.9371) | -5.458 (6.1238) | -6.434 (6.8409) | -6.539 (9.9950)
  Change at Week 4 | -5.722 (8.8627) | -4.889 (7.3568) | -7.948 (7.1614) | -9.819 (11.2688) | -6.560 (8.0631) | -4.754 (7.0439) | -8.050 (6.9054) | -10.433 (11.8548)
  Change at Week 8 | -7.241 (12.4374) | -7.636 (9.0091) | -9.531 (9.5254) | -12.839 (13.1334) | -9.323 (9.2809) | -7.627 (8.9115) | -9.668 (9.4114) | -13.926 (13.7928)
  Change at Week 12 | -7.546 (13.0215) | -10.132 (10.8337) | -12.089 (10.0806) | -13.383 (14.5075) | -9.660 (9.8693) | -10.438 (10.8236) | -12.688 (9.5421) | -14.861 (15.0025)
  Change at Week 16 | -9.294 (13.2176) | -12.043 (10.7104) | -13.809 (9.8357) | -14.152 (14.9552) | -11.853 (9.8578) | -12.565 (10.6334) | -14.322 (9.4641) | -16.617 (14.1166)
  Change at Week 20 | -8.996 (14.7780) | -12.446 (11.0107) | -13.724 (11.8173) | -15.011 (14.9433) | -11.857 (11.8911) | -13.112 (10.9374) | -14.342 (11.5579) | -17.626 (13.9147)
  Change at Week 24 | -8.691 (14.3072) | -12.671 (11.6001) | -14.743 (11.6082) | -14.883 (14.9074) | -11.506 (11.2985) | -13.354 (11.5619) | -15.442 (11.2609) | -17.698 (13.7260)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -13.996 (12.0029) | -14.858 (12.5133) | -16.818 (11.9239) | -18.889 (13.9459)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -15.079 (12.8557) | -15.423 (12.0649) | -15.476 (13.3711) | -18.833 (14.4014)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -14.017 (13.8170) | -14.150 (11.6401) | -17.282 (11.4617) | -20.687 (14.6462)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -14.391 (14.1550) | -14.612 (11.3920) | -17.076 (9.4960) | -19.520 (14.2756)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -13.538 (13.2755) | -14.404 (11.6971) | -16.800 (10.1413) | -20.109 (15.3423)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -13.832 (14.8785) | -14.912 (12.1638) | -16.926 (11.5097) | -19.939 (14.1463)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -13.251 (14.2737) | -14.265 (11.9806) | -16.856 (9.6991) | -19.215 (13.0405)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -14.113 (13.7397) | -14.904 (11.8237) | -16.258 (11.2435) | -20.439 (13.0531)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -14.166 (13.8122) | -15.538 (11.5883) | -16.628 (12.4186) | -20.746 (13.3296)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -14.732 (14.5591) | -15.492 (11.6393) | -15.386 (12.5672) | -20.611 (12.3814)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -15.549 (14.3214) | -14.185 (13.1359) | -16.294 (12.4571) | -21.280 (12.9457)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -14.706 (14.9924) | -14.619 (12.0768) | -16.788 (11.9283) | -20.348 (12.9401)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -14.621 (14.7575) | -14.977 (11.4630) | -17.514 (12.1319) | -20.696 (12.4896)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -14.289 (15.0957) | -15.888 (11.9316) | -17.069 (11.6199) | -20.822 (13.5723)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -14.906 (15.1056) | -15.419 (11.9932) | -17.233 (11.9661) | -20.485 (14.2038)

16. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Values at Each Visit Based on LOCF
Description: The CDAI was calculated from tender joint counts of 28, swollen joint counts of 28, participant's global assessment of disease activity, physician global assessment of disease activity score, and CRP value. Total score ranged between 0-76. CDAI score of 22 or above = high disease activity, a value between 10 and 22 = moderate disease activity and value less than or equal to <=10 = low disease activity, value <=2.8 = disease remission. Higher scores indicated higher disease activity. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
score on a scale
  Baseline | 29.198 (10.1188) | 29.104 (11.3057) | 30.563 (9.3260) | 33.169 (12.0220) | 28.900 (9.9333) | 29.196 (11.7439) | 29.918 (8.2741) | 32.848 (11.4735)
  Change at Week 2 | -5.007 (7.9447) | -5.336 (6.0158) | -6.785 (6.8641) | -6.424 (9.5389) | -5.640 (6.8069) | -5.142 (6.0961) | -6.518 (6.7345) | -6.663 (9.9570)
  Change at Week 4 | -5.787 (8.3763) | -5.093 (6.9306) | -7.983 (7.0449) | -10.152 (10.7576) | -6.421 (7.7106) | -4.904 (6.6827) | -8.080 (6.8543) | -10.713 (11.3327)
  Change at Week 8 | -7.456 (11.9815) | -7.754 (8.3585) | -9.824 (9.4091) | -12.809 (12.4854) | -9.364 (9.0361) | -7.704 (8.2942) | -9.946 (9.3095) | -13.778 (13.1305)
  Change at Week 12 | -7.700 (12.4359) | -9.900 (10.7410) | -12.391 (9.5546) | -13.335 (13.7520) | -9.666 (9.4769) | -10.177 (10.7463) | -13.012 (8.9533) | -14.617 (14.3068)
  Change at Week 16 | -9.469 (12.5253) | -11.786 (10.2476) | -13.698 (9.5039) | -14.243 (14.0490) | -11.853 (9.2509) | -12.273 (10.1616) | -14.220 (9.1180) | -16.541 (13.2391)
  Change at Week 20 | -9.231 (14.0979) | -12.279 (10.3590) | -13.548 (11.4067) | -15.113 (14.3180) | -11.857 (11.3698) | -12.862 (10.2616) | -14.108 (11.1938) | -17.487 (13.3908)
  Change at Week 24 | -9.080 (13.2957) | -12.411 (10.6684) | -14.815 (11.3164) | -15.361 (14.0888) | -11.683 (10.2413) | -13.004 (10.5902) | -15.476 (11.0172) | -18.000 (12.8580)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 28 |  |  |  |  | -13.753 (11.1661) | -14.519 (11.5712) | -16.604 (11.5179) | -18.700 (13.2130)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 32 |  |  |  |  | -14.981 (11.8964) | -15.108 (11.2046) | -15.606 (12.5181) | -18.478 (13.6585)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 36 |  |  |  |  | -13.917 (13.0248) | -14.015 (10.4490) | -17.134 (10.9034) | -20.450 (13.8226)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 40 |  |  |  |  | -14.226 (13.3556) | -14.315 (10.3937) | -16.980 (9.3329) | -19.274 (13.4909)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 44 |  |  |  |  | -13.440 (12.6798) | -14.058 (10.6267) | -17.060 (9.8900) | -19.941 (14.6274)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 48 |  |  |  |  | -13.977 (14.2191) | -14.658 (11.0874) | -16.884 (11.0023) | -19.624 (13.4005)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | -13.577 (13.4474) | -14.031 (10.7633) | -16.764 (9.4282) | -19.076 (12.7465)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 56 |  |  |  |  | -14.019 (12.9269) | -14.462 (10.8608) | -16.228 (10.8175) | -20.167 (12.7089)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 60 |  |  |  |  | -14.032 (12.9707) | -15.400 (10.4881) | -16.592 (11.8366) | -20.354 (12.8739)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 64 |  |  |  |  | -14.687 (13.6997) | -15.150 (10.5316) | -15.924 (11.5956) | -20.215 (12.0216)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 68 |  |  |  |  | -15.291 (13.2786) | -13.958 (12.0080) | -16.422 (11.7994) | -20.917 (12.3462)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 72 |  |  |  |  | -14.536 (13.7461) | -14.346 (10.9159) | -16.828 (11.2797) | -20.063 (12.2151)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | -14.536 (13.4853) | -14.600 (10.4240) | -17.556 (11.5861) | -20.289 (11.8557)
  Change at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 80 |  |  |  |  | -14.091 (14.0501) | -15.565 (10.7890) | -17.090 (11.0248) | -20.420 (12.9597)
  Change at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 84 |  |  |  |  | -14.679 (13.9556) | -15.031 (10.8769) | -17.344 (11.2309) | -20.139 (13.4967)

17. Secondary Outcome: Number of Participants With a European League Against Rheumatism (EULAR) Good, Moderate or No Response Using DAS28-ESR at Each Visit Based on NRI
Description: The Disease Activity Score Based on 28-joints Count based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 <=3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to <=5.1 or change from baseline >0.6 to <=1.2 with DAS28 <=5.1; non-responders: change from baseline <=0.6 or change from baseline >0.6 and <=1.2 with DAS28 >5.1. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: Treatment Phase: Weeks 2, 4, 8, 12, 16, 20, and 24; Extension Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, and 84
Population: FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given time points. Missing data was imputed using NRI imputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
Participants
  EULAR response at Week 2: number analyzed (Participants) | 53 | 28 | 54 | 53 | 46 | 26 | 50 | 45
  EULAR response at Week 2: Good response | 3 | 1 | 2 | 0 | 3 | 0 | 1 | 0
  EULAR response at Week 2: Moderate response | 12 | 6 | 13 | 11 | 11 | 9 | 14 | 10
  EULAR response at Week 2: No response | 38 | 21 | 39 | 42 | 32 | 17 | 35 | 35
  EULAR response at Week 4: Good response | 2 | 0 | 1 | 2 | 2 | 0 | 1 | 2
  EULAR response at Week 4: Moderate response | 15 | 9 | 22 | 20 | 14 | 8 | 21 | 18
  EULAR response at Week 4: No response | 37 | 19 | 31 | 32 | 31 | 18 | 28 | 26
  EULAR response at Week 8: Good response | 5 | 1 | 4 | 7 | 5 | 1 | 3 | 7
  EULAR response at Week 8: Moderate response | 19 | 13 | 26 | 28 | 17 | 12 | 26 | 24
  EULAR response at Week 8: No response | 30 | 14 | 24 | 19 | 25 | 13 | 21 | 15
  EULAR response at Week 12: Good response | 7 | 3 | 10 | 11 | 7 | 3 | 9 | 11
  EULAR response at Week 12: Moderate response | 18 | 11 | 26 | 19 | 16 | 10 | 26 | 19
  EULAR response at Week 12: No response | 29 | 14 | 18 | 24 | 24 | 13 | 15 | 16
  EULAR response at Week 16: Good response | 10 | 5 | 10 | 9 | 10 | 5 | 10 | 9
  EULAR response at Week 16: Moderate response | 22 | 11 | 29 | 24 | 21 | 10 | 29 | 23
  EULAR response at Week 16: No response | 22 | 12 | 15 | 21 | 16 | 11 | 11 | 14
  EULAR response at Week 20: Good response | 6 | 4 | 13 | 13 | 6 | 4 | 13 | 13
  EULAR response at Week 20: Moderate response | 20 | 15 | 23 | 23 | 20 | 14 | 23 | 23
  EULAR response at Week 20: No response | 28 | 9 | 18 | 18 | 21 | 8 | 14 | 10
  EULAR response at Week 24: Good response | 7 | 4 | 10 | 13 | 7 | 4 | 10 | 13
  EULAR response at Week 24: Moderate response | 19 | 11 | 27 | 21 | 19 | 11 | 27 | 21
  EULAR response at Week 24: No response | 28 | 13 | 17 | 20 | 21 | 11 | 13 | 12
  EULAR response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 28: Good response |  |  |  |  | 11 | 6 | 12 | 13
  EULAR response at Week 28: Moderate response |  |  |  |  | 22 | 10 | 29 | 23
  EULAR response at Week 28: No response |  |  |  |  | 14 | 10 | 9 | 10
  EULAR response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 32: Good response |  |  |  |  | 12 | 5 | 13 | 12
  EULAR response at Week 32: Moderate response |  |  |  |  | 19 | 13 | 26 | 22
  EULAR response at Week 32: No response |  |  |  |  | 16 | 8 | 11 | 12
  EULAR response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 36: Good response |  |  |  |  | 11 | 4 | 12 | 14
  EULAR response at Week 36: Moderate response |  |  |  |  | 25 | 11 | 29 | 22
  EULAR response at Week 36: No response |  |  |  |  | 11 | 11 | 9 | 10
  EULAR response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 40: Good response |  |  |  |  | 12 | 5 | 15 | 13
  EULAR response at Week 40: Moderate response |  |  |  |  | 19 | 9 | 24 | 21
  EULAR response at Week 40: No response |  |  |  |  | 16 | 12 | 11 | 12
  EULAR response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 44: Good response |  |  |  |  | 12 | 5 | 15 | 13
  EULAR response at Week 44: Moderate response |  |  |  |  | 19 | 9 | 24 | 22
  EULAR response at Week 44: No response |  |  |  |  | 16 | 12 | 11 | 11
  EULAR response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 48: Good response |  |  |  |  | 11 | 7 | 14 | 14
  EULAR response at Week 48: Moderate response |  |  |  |  | 23 | 7 | 23 | 20
  EULAR response at Week 48: No response |  |  |  |  | 13 | 12 | 13 | 12
  EULAR response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 52: Good response |  |  |  |  | 14 | 6 | 12 | 16
  EULAR response at Week 52: Moderate response |  |  |  |  | 15 | 8 | 22 | 18
  EULAR response at Week 52: No response |  |  |  |  | 18 | 12 | 16 | 12
  EULAR response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 56: Good response |  |  |  |  | 15 | 6 | 9 | 14
  EULAR response at Week 56: Moderate response |  |  |  |  | 16 | 10 | 27 | 23
  EULAR response at Week 56: No response |  |  |  |  | 16 | 10 | 14 | 9
  EULAR response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 60: Good response |  |  |  |  | 14 | 7 | 17 | 15
  EULAR response at Week 60: Moderate response |  |  |  |  | 17 | 9 | 17 | 19
  EULAR response at Week 60: No response |  |  |  |  | 16 | 10 | 16 | 12
  EULAR response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 64: Good response |  |  |  |  | 14 | 8 | 13 | 15
  EULAR response at Week 64: Moderate response |  |  |  |  | 18 | 7 | 21 | 23
  EULAR response at Week 64: No response |  |  |  |  | 15 | 11 | 16 | 8
  EULAR response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 68: Good response |  |  |  |  | 15 | 6 | 15 | 17
  EULAR response at Week 68: Moderate response |  |  |  |  | 17 | 8 | 19 | 20
  EULAR response at Week 68: No response |  |  |  |  | 15 | 12 | 16 | 9
  EULAR response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 72: Good response |  |  |  |  | 11 | 4 | 13 | 18
  EULAR response at Week 72: Moderate response |  |  |  |  | 18 | 11 | 19 | 16
  EULAR response at Week 72: No response |  |  |  |  | 18 | 11 | 18 | 12
  EULAR response at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 76: Good response |  |  |  |  | 11 | 6 | 16 | 18
  EULAR response at Week 76: Moderate response |  |  |  |  | 19 | 9 | 16 | 19
  EULAR response at Week 76: No response |  |  |  |  | 17 | 11 | 18 | 9
  EULAR response at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 80: Good response |  |  |  |  | 13 | 5 | 12 | 19
  EULAR response at Week 80: Moderate response |  |  |  |  | 16 | 11 | 21 | 16
  EULAR response at Week 80: No response |  |  |  |  | 18 | 10 | 17 | 11
  EULAR response at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 84: Good response |  |  |  |  | 12 | 8 | 13 | 17
  EULAR response at Week 84: Moderate response |  |  |  |  | 21 | 7 | 21 | 17
  EULAR response at Week 84: No response |  |  |  |  | 14 | 11 | 16 | 12

18. Secondary Outcome: Number of Participants With a EULAR Good or Moderate Response Using DAS28-CRP at Each Visit Based on NRI
Description: as for outcome 17
Time Frame: as for outcome 17
Population: FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given time points. Missing data was imputed using NRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
Participants
  EULAR response at Week 2: Good response | 3 | 1 | 2 | 0 | 3 | 1 | 2 | 0
  EULAR response at Week 2: Moderate response | 11 | 6 | 13 | 12 | 10 | 5 | 10 | 11
  EULAR response at Week 2: No response | 40 | 21 | 39 | 42 | 34 | 20 | 38 | 35
  EULAR response at Week 4: Good response | 2 | 0 | 3 | 3 | 2 | 0 | 3 | 3
  EULAR response at Week 4: Moderate response | 13 | 8 | 17 | 18 | 12 | 7 | 16 | 17
  EULAR response at Week 4: No response | 39 | 20 | 34 | 33 | 33 | 19 | 31 | 26
  EULAR response at Week 8: Good response | 5 | 1 | 8 | 6 | 5 | 1 | 7 | 6
  EULAR response at Week 8: Moderate response | 14 | 12 | 19 | 23 | 13 | 11 | 19 | 21
  EULAR response at Week 8: No response | 35 | 15 | 27 | 25 | 29 | 14 | 24 | 19
  EULAR response at Week 12: Good response | 7 | 6 | 14 | 8 | 7 | 6 | 13 | 8
  EULAR response at Week 12: Moderate response | 16 | 8 | 17 | 21 | 15 | 7 | 17 | 21
  EULAR response at Week 12: No response | 31 | 14 | 23 | 25 | 25 | 13 | 20 | 17
  EULAR response at Week 16: Good response | 9 | 5 | 12 | 12 | 9 | 5 | 12 | 12
  EULAR response at Week 16: Moderate response | 20 | 10 | 23 | 18 | 19 | 9 | 23 | 16
  EULAR response at Week 16: No response | 25 | 13 | 19 | 24 | 19 | 12 | 15 | 18
  EULAR response at Week 20: Good response | 8 | 5 | 15 | 15 | 8 | 5 | 15 | 15
  EULAR response at Week 20: Moderate response | 17 | 12 | 21 | 17 | 17 | 12 | 21 | 17
  EULAR response at Week 20: No response | 29 | 11 | 18 | 22 | 22 | 9 | 14 | 14
  EULAR response at Week 24: Good response | 8 | 7 | 14 | 14 | 8 | 7 | 14 | 14
  EULAR response at Week 24: Moderate response | 17 | 6 | 18 | 17 | 17 | 6 | 18 | 17
  EULAR response at Week 24: No response | 29 | 15 | 22 | 23 | 22 | 13 | 18 | 15
  EULAR response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 28: Good response |  |  |  |  | 9 | 5 | 16 | 15
  EULAR response at Week 28: Moderate response |  |  |  |  | 23 | 12 | 21 | 17
  EULAR response at Week 28: No response |  |  |  |  | 15 | 9 | 13 | 14
  EULAR response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 32: Good response |  |  |  |  | 13 | 5 | 17 | 16
  EULAR response at Week 32: Moderate response |  |  |  |  | 16 | 14 | 19 | 15
  EULAR response at Week 32: No response |  |  |  |  | 18 | 7 | 14 | 15
  EULAR response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 36: Good response |  |  |  |  | 12 | 5 | 16 | 17
  EULAR response at Week 36: Moderate response |  |  |  |  | 23 | 11 | 22 | 20
  EULAR response at Week 36: No response |  |  |  |  | 12 | 10 | 12 | 9
  EULAR response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 40: Good response |  |  |  |  | 11 | 5 | 15 | 14
  EULAR response at Week 40: Moderate response |  |  |  |  | 16 | 10 | 22 | 21
  EULAR response at Week 40: No response |  |  |  |  | 20 | 11 | 13 | 11
  EULAR response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 44: Good response |  |  |  |  | 11 | 5 | 16 | 16
  EULAR response at Week 44: Moderate response |  |  |  |  | 19 | 9 | 20 | 16
  EULAR response at Week 44: No response |  |  |  |  | 17 | 12 | 14 | 14
  EULAR response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 48: Good response |  |  |  |  | 11 | 7 | 17 | 17
  EULAR response at Week 48: Moderate response |  |  |  |  | 21 | 8 | 18 | 14
  EULAR response at Week 48: No response |  |  |  |  | 15 | 11 | 15 | 15
  EULAR response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 52: Good response |  |  |  |  | 16 | 7 | 12 | 18
  EULAR response at Week 52: Moderate response |  |  |  |  | 11 | 6 | 21 | 14
  EULAR response at Week 52: No response |  |  |  |  | 20 | 13 | 17 | 14
  EULAR response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 56: Good response |  |  |  |  | 16 | 6 | 15 | 21
  EULAR response at Week 56: Moderate response |  |  |  |  | 13 | 11 | 19 | 14
  EULAR response at Week 56: No response |  |  |  |  | 18 | 9 | 16 | 11
  EULAR response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 60: Good response |  |  |  |  | 15 | 8 | 16 | 18
  EULAR response at Week 60: Moderate response |  |  |  |  | 15 | 9 | 18 | 16
  EULAR response at Week 60: No response |  |  |  |  | 17 | 9 | 16 | 12
  EULAR response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 64: Good response |  |  |  |  | 12 | 7 | 15 | 19
  EULAR response at Week 64: Moderate response |  |  |  |  | 18 | 9 | 18 | 17
  EULAR response at Week 64: No response |  |  |  |  | 17 | 10 | 17 | 10
  EULAR response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 68: Good response |  |  |  |  | 16 | 7 | 17 | 18
  EULAR response at Week 68: Moderate response |  |  |  |  | 17 | 7 | 17 | 19
  EULAR response at Week 68: No response |  |  |  |  | 14 | 12 | 16 | 9
  EULAR response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 72: Good response |  |  |  |  | 12 | 7 | 19 | 18
  EULAR response at Week 72: Moderate response |  |  |  |  | 16 | 8 | 12 | 15
  EULAR response at Week 72: No response |  |  |  |  | 19 | 11 | 19 | 13
  EULAR response at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 76: Good response |  |  |  |  | 15 | 7 | 18 | 20
  EULAR response at Week 76: Moderate response |  |  |  |  | 15 | 9 | 15 | 15
  EULAR response at Week 76: No response |  |  |  |  | 17 | 10 | 17 | 11
  EULAR response at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 80: Good response |  |  |  |  | 15 | 8 | 14 | 22
  EULAR response at Week 80: Moderate response |  |  |  |  | 14 | 7 | 19 | 12
  EULAR response at Week 80: No response |  |  |  |  | 18 | 11 | 17 | 12
  EULAR response at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  EULAR response at Week 84: Good response |  |  |  |  | 15 | 8 | 19 | 22
  EULAR response at Week 84: Moderate response |  |  |  |  | 16 | 7 | 15 | 12
  EULAR response at Week 84: No response |  |  |  |  | 16 | 11 | 16 | 12

19. Secondary Outcome: Percentage of Participants Who Achieved SDAI Remission at Each Visit Based on NRI
Description: The SDAI was calculated from tender joint counts of 28, swollen joint counts of 28, participant's global assessment of disease activity, physician global assessment of disease activity score, and CRP value. Total score ranged between 0-86. SDAI score of 26 or above = high disease activity, a value between 11 and 26 = moderate disease activity and value <=11 = low disease activity. Higher scores indicated higher disease activity. SDAI Remission was defined as SDAI score <=3.3. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: Treatment Phase: Weeks 2, 4, 8, 12, 16, 20, and 24; Extension Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, and 104
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
percentage of participants
  Remission at Week 2 | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 2.1 [0.00 to 6.25] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 4 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 2.0 [0.00 to 5.88] | 0.0 [0.00 to 0.00]
  Remission at Week 8 | 0.0 [0.00 to 0.00] | 3.6 [0.00 to 10.45] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 3.8 [0.00 to 11.24] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 12 | 1.9 [0.00 to 5.45] | 10.7 [0.00 to 22.17] | 3.7 [0.00 to 8.74] | 1.9 [0.00 to 5.45] | 2.1 [0.00 to 6.25] | 11.5 [0.00 to 23.82] | 4.0 [0.00 to 9.43] | 2.2 [0.00 to 6.39]
  Remission at Week 16 | 3.7 [0.00 to 8.74] | 10.7 [0.00 to 22.17] | 5.6 [0.00 to 11.67] | 3.7 [0.00 to 8.74] | 4.3 [0.00 to 10.03] | 11.5 [0.00 to 23.82] | 6.0 [0.00 to 12.58] | 4.3 [0.00 to 10.24]
  Remission at Week 20 | 7.4 [0.42 to 14.39] | 14.3 [1.32 to 27.25] | 7.4 [0.42 to 14.39] | 9.3 [1.53 to 16.99] | 8.5 [0.53 to 16.49] | 15.4 [1.52 to 29.25] | 8.0 [0.48 to 15.52] | 10.9 [1.87 to 19.86]
  Remission at Week 24 | 5.6 [0.00 to 11.67] | 7.1 [0.00 to 16.68] | 7.4 [0.42 to 14.39] | 11.1 [2.73 to 19.49] | 6.4 [0.00 to 13.37] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 13.0 [3.31 to 22.78]
  Remission at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 28 |  |  |  |  | 6.4 [0.00 to 13.37] | 11.5 [0.00 to 23.82] | 10.0 [1.68 to 18.32] | 10.9 [1.87 to 19.86]
  Remission at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 32 |  |  |  |  | 8.5 [0.53 to 16.49] | 11.5 [0.00 to 23.82] | 10.0 [1.68 to 18.32] | 13.0 [3.31 to 22.78]
  Remission at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 36 |  |  |  |  | 8.5 [0.53 to 16.49] | 7.7 [0.00 to 17.93] | 14.0 [4.38 to 23.62] | 13.0 [3.31 to 22.78]
  Remission at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 40 |  |  |  |  | 12.8 [3.23 to 22.31] | 7.7 [0.00 to 17.93] | 12.0 [2.99 to 21.01] | 15.2 [4.84 to 25.60]
  Remission at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 44 |  |  |  |  | 10.6 [1.82 to 19.45] | 11.5 [0.00 to 23.82] | 16.0 [5.84 to 26.16] | 15.2 [4.84 to 25.60]
  Remission at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 48 |  |  |  |  | 17.0 [6.28 to 27.77] | 19.2 [4.08 to 34.38] | 12.0 [2.99 to 21.01] | 21.7 [9.82 to 33.66]
  Remission at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 52 |  |  |  |  | 17.0 [6.28 to 27.77] | 15.4 [1.52 to 29.25] | 10.0 [1.68 to 18.32] | 13.0 [3.31 to 22.78]
  Remission at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 56 |  |  |  |  | 14.9 [4.72 to 25.07] | 15.4 [1.52 to 29.25] | 6.0 [0.00 to 12.58] | 17.4 [6.44 to 28.34]
  Remission at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 60 |  |  |  |  | 12.8 [3.23 to 22.31] | 19.2 [4.08 to 34.38] | 16.0 [5.84 to 26.16] | 13.0 [3.31 to 22.78]
  Remission at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 64 |  |  |  |  | 10.6 [1.82 to 19.45] | 19.2 [4.08 to 34.38] | 12.0 [2.99 to 21.01] | 10.9 [1.87 to 19.86]
  Remission at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 68 |  |  |  |  | 19.1 [7.90 to 30.40] | 23.1 [6.88 to 39.27] | 8.0 [0.48 to 15.52] | 17.4 [6.44 to 28.34]
  Remission at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 72 |  |  |  |  | 10.6 [1.82 to 19.45] | 19.2 [4.08 to 34.38] | 14.0 [4.38 to 23.62] | 19.6 [8.10 to 31.03]
  Remission at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 76 |  |  |  |  | 10.6 [1.82 to 19.45] | 19.2 [4.08 to 34.38] | 6.0 [0.00 to 12.58] | 17.4 [6.44 to 28.34]
  Remission at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 80 |  |  |  |  | 19.1 [7.90 to 30.40] | 15.4 [1.52 to 29.25] | 4.0 [0.00 to 9.43] | 26.1 [13.40 to 38.78]
  Remission at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 84 |  |  |  |  | 17.0 [6.28 to 27.77] | 23.1 [6.88 to 39.27] | 12.0 [2.99 to 21.01] | 23.9 [11.59 to 36.24]

20. Secondary Outcome: Percentage of Participants Who Achieved CDAI Remission at Each Visit Based on NRI
Description: The CDAI was calculated from tender joint counts of 28, swollen joint counts of 28, participant's global assessment of disease activity, physician global assessment of disease activity score, and CRP value. Total score ranged between 0-76. CDAI score of 22 or above = high disease activity, a value between 10 and 22 = moderate disease activity and value less than or equal to <=10 = low disease activity. Higher scores indicated higher disease activity. CDAI Remission was defined as CDAI score <=2.8. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: Treatment Phase: Weeks 2, 4, 8, 12, 16, 20, and 24; Extension Phase: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, and 84
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
percentage of participants
  Remission at Week 2 | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 2.1 [0.00 to 6.25] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 4 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 8 | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 2.1 [0.00 to 6.25] | 0.0 [0.00 to 0.00] | 2.0 [0.00 to 5.88] | 0.0 [0.00 to 0.00]
  Remission at Week 12 | 1.9 [0.00 to 5.45] | 7.1 [0.00 to 16.68] | 3.7 [0.00 to 8.74] | 1.9 [0.00 to 5.45] | 2.1 [0.00 to 6.25] | 7.7 [0.00 to 17.93] | 4.0 [0.00 to 9.43] | 2.2 [0.00 to 6.39]
  Remission at Week 16 | 3.7 [0.00 to 8.74] | 10.7 [0.00 to 22.17] | 5.6 [0.00 to 11.67] | 3.7 [0.00 to 8.74] | 4.3 [0.00 to 10.03] | 11.5 [0.00 to 23.82] | 6.0 [0.00 to 12.58] | 4.3 [0.00 to 10.24]
  Remission at Week 20 | 7.4 [0.42 to 14.39] | 10.7 [0.00 to 22.17] | 7.4 [0.42 to 14.39] | 9.3 [1.53 to 16.99] | 8.5 [0.53 to 16.49] | 11.5 [0.00 to 23.82] | 8.0 [0.48 to 15.52] | 10.9 [1.87 to 19.86]
  Remission at Week 24 | 5.6 [0.00 to 11.67] | 7.1 [0.00 to 16.68] | 7.4 [0.42 to 14.39] | 9.3 [1.53 to 16.99] | 6.4 [0.00 to 13.37] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 10.9 [1.87 to 19.86]
  Remission at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 28 |  |  |  |  | 8.5 [0.53 to 16.49] | 11.5 [0.00 to 23.82] | 8.0 [0.48 to 15.52] | 10.9 [1.87 to 19.86]
  Remission at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 32 |  |  |  |  | 6.4 [0.00 to 13.37] | 7.7 [0.00 to 17.93] | 10.0 [1.68 to 18.32] | 13.0 [3.31 to 22.78]
  Remission at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 36 |  |  |  |  | 6.4 [0.00 to 13.37] | 0.0 [0.00 to 0.00] | 12.0 [2.99 to 21.01] | 15.2 [4.84 to 25.60]
  Remission at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 40 |  |  |  |  | 8.5 [0.53 to 16.49] | 3.8 [0.00 to 11.24] | 8.0 [0.48 to 15.52] | 13.0 [3.31 to 22.78]
  Remission at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 44 |  |  |  |  | 8.5 [0.53 to 16.49] | 7.7 [0.00 to 17.93] | 16.0 [5.84 to 26.16] | 15.2 [4.84 to 25.60]
  Remission at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 48 |  |  |  |  | 17.0 [6.28 to 27.77] | 11.5 [0.00 to 23.82] | 12.0 [2.99 to 21.01] | 19.6 [8.10 to 31.03]
  Remission at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 52 |  |  |  |  | 19.1 [7.90 to 30.40] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 13.0 [3.31 to 22.78]
  Remission at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 56 |  |  |  |  | 10.6 [1.82 to 19.45] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 17.4 [6.44 to 28.34]
  Remission at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 60 |  |  |  |  | 12.8 [3.23 to 22.31] | 11.5 [0.00 to 23.82] | 14.0 [4.38 to 23.62] | 13.0 [3.31 to 22.78]
  Remission at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 64 |  |  |  |  | 8.5 [0.53 to 16.49] | 19.2 [4.08 to 34.38] | 12.0 [2.99 to 21.01] | 10.9 [1.87 to 19.86]
  Remission at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 68 |  |  |  |  | 19.1 [7.90 to 30.40] | 19.2 [4.08 to 34.38] | 8.0 [0.48 to 15.52] | 19.6 [8.10 to 31.03]
  Remission at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 72 |  |  |  |  | 10.6 [1.82 to 19.45] | 15.4 [1.52 to 29.25] | 12.0 [2.99 to 21.01] | 17.4 [6.44 to 28.34]
  Remission at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 76 |  |  |  |  | 10.6 [1.82 to 19.45] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 19.6 [8.10 to 31.03]
  Remission at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 80 |  |  |  |  | 19.1 [7.90 to 30.40] | 15.4 [1.52 to 29.25] | 2.0 [0.00 to 5.88] | 23.9 [11.59 to 36.24]
  Remission at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 84 |  |  |  |  | 14.9 [4.72 to 25.07] | 23.1 [6.88 to 39.27] | 10.0 [1.68 to 18.32] | 23.9 [11.59 to 36.24]

21. Secondary Outcome: Percentage of Participants Who Achieved Boolean Remission at Each Visit Based on NRI
Description: Boolean remission criteria was defined as: tender joint count 68 <=1; swollen joint count 68 <=1; CRP <=1 mg/dL; and disease activity assessments VAS (mm) by participants <=1. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: as for outcome 20
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
percentage of participants
  Remission at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 4 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.9 [0.00 to 5.45] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 2.0 [0.00 to 5.88] | 0.0 [0.00 to 0.00]
  Remission at Week 8 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 12 | 1.9 [0.00 to 5.45] | 3.6 [0.00 to 10.45] | 3.7 [0.00 to 8.74] | 3.7 [0.00 to 8.74] | 2.1 [0.00 to 6.25] | 3.8 [0.00 to 11.24] | 4.0 [0.00 to 9.43] | 4.3 [0.00 to 10.24]
  Remission at Week 16 | 1.9 [0.00 to 5.45] | 7.1 [0.00 to 16.68] | 3.7 [0.00 to 8.74] | 3.7 [0.00 to 8.74] | 2.1 [0.00 to 6.25] | 7.7 [0.00 to 17.93] | 4.0 [0.00 to 9.43] | 4.3 [0.00 to 10.24]
  Remission at Week 20 | 0.0 [0.00 to 0.00] | 3.6 [0.00 to 10.45] | 3.7 [0.00 to 8.74] | 9.3 [1.53 to 16.99] | 0.0 [0.00 to 0.00] | 3.8 [0.00 to 11.24] | 4.0 [0.00 to 9.43] | 10.9 [1.87 to 19.86]
  Remission at Week 24 | 1.9 [0.00 to 5.45] | 3.6 [0.00 to 10.45] | 5.6 [0.00 to 11.67] | 5.6 [0.00 to 11.67] | 2.1 [0.00 to 6.25] | 3.8 [0.00 to 11.24] | 6.0 [0.00 to 12.58] | 6.5 [0.00 to 13.66]
  Remission at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 28 |  |  |  |  | 4.3 [0.00 to 10.03] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 6.5 [0.00 to 13.66]
  Remission at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 32 |  |  |  |  | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 17.93] | 6.0 [0.00 to 12.58] | 8.7 [0.55 to 16.84]
  Remission at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 36 |  |  |  |  | 2.1 [0.00 to 6.25] | 7.7 [0.00 to 17.93] | 10.0 [1.68 to 18.32] | 8.7 [0.55 to 16.84]
  Remission at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 40 |  |  |  |  | 4.3 [0.00 to 10.03] | 11.5 [0.00 to 23.82] | 4.0 [0.00 to 9.43] | 8.7 [0.55 to 16.84]
  Remission at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 44 |  |  |  |  | 2.1 [0.00 to 6.25] | 7.7 [0.00 to 17.93] | 14.0 [4.38 to 23.62] | 8.7 [0.55 to 16.84]
  Remission at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 48 |  |  |  |  | 4.3 [0.00 to 10.03] | 7.7 [0.00 to 17.93] | 10.0 [1.68 to 18.32] | 15.2 [4.84 to 25.60]
  Remission at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 52 |  |  |  |  | 6.4 [0.00 to 13.37] | 3.8 [0.00 to 11.24] | 6.0 [0.00 to 12.58] | 8.7 [0.55 to 16.84]
  Remission at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 56 |  |  |  |  | 4.3 [0.00 to 10.03] | 7.7 [0.00 to 17.93] | 6.0 [0.00 to 12.58] | 10.9 [1.87 to 19.86]
  Remission at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 60 |  |  |  |  | 6.4 [0.00 to 13.37] | 7.7 [0.00 to 17.93] | 10.0 [1.68 to 18.32] | 6.5 [0.00 to 13.66]
  Remission at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 64 |  |  |  |  | 10.6 [1.82 to 19.45] | 7.7 [0.00 to 17.93] | 6.0 [0.00 to 12.58] | 8.7 [0.55 to 16.84]
  Remission at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 68 |  |  |  |  | 10.6 [1.82 to 19.45] | 11.5 [0.00 to 23.82] | 6.0 [0.00 to 12.58] | 8.7 [0.55 to 16.84]
  Remission at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 72 |  |  |  |  | 6.4 [0.00 to 13.37] | 7.7 [0.00 to 17.93] | 8.0 [0.48 to 15.52] | 15.2 [4.84 to 25.60]
  Remission at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 76 |  |  |  |  | 2.1 [0.00 to 6.25] | 11.5 [0.00 to 23.82] | 4.0 [0.00 to 9.43] | 15.2 [4.84 to 25.60]
  Remission at Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 80 |  |  |  |  | 8.5 [0.53 to 16.49] | 11.5 [0.00 to 23.82] | 6.0 [0.00 to 12.58] | 19.6 [8.10 to 31.03]
  Remission at Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Remission at Week 84 |  |  |  |  | 8.5 [0.53 to 16.49] | 11.5 [0.00 to 23.82] | 6.0 [0.00 to 12.58] | 19.6 [8.10 to 31.03]

22. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Each Visit Based on Observed Cases (OC)
Description: The mTSS was a measure of change in joint health. X-rays of hands, wrists, and feet (including distal interphalangeal joints) were obtained. Totals for hands and feet for erosion scores (range 0 to 320) and joint space narrowing scores (range 0 to 208) were calculated and added to obtain the mTSS (range = 0 [normal] to 528 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening; no progression was defined as a change of <=0.5. Data reported for the Extension Phase from Baseline and Week 24, is the same data for the Treatment Phase, but excluding the participants who did not gave consent to participate in Extension Phase.
Time Frame: Treatment Phase: Baseline and Week 24; Extension Phase: Baseline, Weeks 24, 52, 76, and 104
Population: FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given time points. Missing data was imputed using OC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
Number analyzed (Participants) | 54 | 28 | 54 | 54 | 47 | 26 | 50 | 46
units on a scale
  Baseline | 27.20 (46.948) | 30.00 (36.582) | 37.55 (56.095) | 27.64 (40.621) | 17.08 (25.897) | 29.11 (34.551) | 31.61 (47.092) | 26.19 (35.524)
  Change at Week 24 | 1.31 (2.639) | 2.54 (4.768) | 1.82 (4.075) | 1.34 (3.106) | 1.01 (1.929) | 1.20 (3.092) | 0.95 (3.392) | 0.49 (1.438)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 52 |  |  |  |  | 2.37 (4.302) | 3.11 (4.711) | 3.35 (10.366) | 1.33 (3.559)
  Change at Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 76 |  |  |  |  | 3.00 (5.931) | 3.61 (5.631) | 3.96 (14.378) | 1.63 (3.992)
  Change at Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0 | 47 | 26 | 50 | 46
  Change at Week 104 |  |  |  |  | 3.49 (6.643) | 4.02 (5.598) | 4.70 (17.549) | 1.57 (3.885)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 104 Weeks (Treatment Phase: From the first dose of study drug till Week 24; Extension Phase: Post Week 24 till Week 104])
Arm/Group | Treatment Phase: Placebo | Treatment Phase: E6011 100 mg | Treatment Phase: E6011 200 mg | Treatment Phase: E6011 400/200 mg | Extension Phase: Placebo | Extension Phase: E6011 100 mg | Extension Phase: E6011 200 mg | Extension Phase: E6011 400/200 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/28 | 0/54 | 0/54 | 0/47 | 0/26 | 0/50 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/28 | 2/54 | 3/54 | 4/47 | 1/26 | 7/50 | 6/46
Other Adverse Events (participants affected / at risk) | 34/54 | 19/28 | 38/54 | 43/54 | 46/47 | 26/26 | 50/50 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: Placebo (N=54) | Treatment Phase: E6011 100 mg (N=28) | Treatment Phase: E6011 200 mg (N=54) | Treatment Phase: E6011 400/200 mg (N=54) | Extension Phase: Placebo (N=47) | Extension Phase: E6011 100 mg (N=26) | Extension Phase: E6011 200 mg (N=50) | Extension Phase: E6011 400/200 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular stent restenosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase: Placebo (N=54) | Treatment Phase: E6011 100 mg (N=28) | Treatment Phase: E6011 200 mg (N=54) | Treatment Phase: E6011 400/200 mg (N=54) | Extension Phase: Placebo (N=47) | Extension Phase: E6011 100 mg (N=26) | Extension Phase: E6011 200 mg (N=50) | Extension Phase: E6011 400/200 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 3 | 3 | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Dry eye (Eye disorders) | 2 | 0 | 0 | 2 | 2 | 0 | 2 | 2
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 5 | 3 | 2 | 3 | 7
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 5
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 4 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 2 | 3 | 3 | 2
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1
Injection site erythema (General disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 3 | 3
Injection site reaction (General disorders) | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2
Injection site pruritus (General disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 2 | 2 | 1 | 0 | 5 | 2
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 16 | 7 | 10 | 18 | 28 | 15 | 30 | 28
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4 | 2 | 4 | 3 | 7 | 4
Bronchitis (Infections and infestations) | 1 | 2 | 1 | 3 | 4 | 3 | 3 | 5
Pharyngitis (Infections and infestations) | 2 | 0 | 3 | 2 | 4 | 2 | 4 | 4
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 4 | 2 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 6 | 2 | 2 | 2
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 1 | 3 | 3
Gingival abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 2 | 2 | 2 | 5 | 4
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Cell marker increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Procalcitonin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 2 | 4 | 2 | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 5 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Vagus nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 1 | 3 | 0 | 1 | 2
Somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 4 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3 | 2 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 2 | 1 | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 2 | 4 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 4 | 3 | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukoplakia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bacterial vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tracheobronchitis mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Human chorionic gonadotropin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mycobacterium tuberculosis complex test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Double stranded DNA antibody positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyslalia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bulimia nervosa (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Internal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02960438/Prot_000.pdf
  • Statistical Analysis Plan: Treatment Phase (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT02960438/SAP_001.pdf
  • Statistical Analysis Plan: Extension Phase (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT02960438/SAP_002.pdf